CLINICAL TRIAL: NCT02939131
Title: IMPAACT 2002: Combined Cognitive Behavioral Therapy and a Medication Management Algorithm for Treatment of Depression Among Youth Living With HIV in the United States
Brief Title: IMPAACT 2002: Cognitive Behavioral Therapy and Medication Management for Treatment of Depression in US Youth With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2002; UM1AI068632 (NIH); UM1AI068616 (NIH); UM1AI106716 (NIH)
Record Dates: First submitted 2016-10-07; First posted 2016-10-19 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: HIV; Depression
Keywords: Cognitive Behavioral Therapy; Medication Management
MeSH Terms: conditions — Depression | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMB-R (Experimental): Health and Wellness Cognitive Behavioral Therapy and Medication Management (COMB-R) intervention
  Interventions: Behavioral: Health and Wellness Combined Cognitive Behavioral Therapy and a Medication Management Algorithm
- Enhanced Standard of Care (Active Comparator): Enhanced Standard of Care (ESC)
  Interventions: Behavioral: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Health and Wellness Combined Cognitive Behavioral Therapy and a Medication Management Algorithm — Behavioral therapy based on a manualized approach developed specifically for youth living with both HIV and depression, using problem-solving, motivational interviewing and cognitive-behavioral strategies to decrease adherence obstacles and increase wellness. The medication management algorithm includes guidance for clinicians on strategies and tactics to treat depression in this population, including factors to consider when deciding on treatments (i.e., drug-drug interactions, side effects).
  Arms: COMB-R
Behavioral: Enhanced Standard of Care — Ongoing psychopharmacological and psychosocial counseling and treatment for depression at HIV clinical treatment centers enhanced by providing clinicians with up-to-date information and didactic training on current principles for use of medication and psychotherapy in the treatment of depression.
  Arms: Enhanced Standard of Care

SUMMARY:
IMPAACT 2002 is a prospective, multi-site, two-arm, cluster-randomized study to evaluate whether a health and wellness Cognitive Behavioral Therapy and Medication Management (COMB-R) intervention for depression demonstrates improved depression and medical outcomes for HIV-infected youth in the United States (US) compared to enhanced standard care (ESC).

DETAILED DESCRIPTION:
IMPAACT 2002 was a prospective, multi-site, two-arm, cluster-randomized study that evaluated whether a health and wellness Cognitive Behavioral Therapy and Medication Management (COMB-R) intervention for depression demonstrated improved depression outcomes (e.g., decreased depressive symptoms and greater remission and response rates) and medical outcomes (e.g., increased cluster of differentiation 4 (CD4) T-cell count, decreased HIV RNA level) among HIV-infected youth in the US compared to enhanced standard care (ESC). Sites were randomized to either the COMB-R intervention or the ESC control arm. Youth enrolled in the study attended a Screening/Entry Visit and study visits at Weeks 1, 6, 12, and 24. They had two additional follow-up visits at Weeks 36 and 48 for the study team to evaluate if observed effects of the intervention were maintained. The intervention was a treatment for depression that included a manualized Health and Wellness Cognitive Behavioral Therapy and an algorithm-driven Medication Management designed to address the unique challenges faced by this population.

ELIGIBILITY:
Inclusion Criteria:

* Receiving mental health or HIV-related care at participating US IMPAACT site
* Confirmed HIV-1 Infection
* Aware of his or her HIV infection
* Per clinician assessment, primary diagnosis of nonpsychotic depression, including Major Depressive Disorder, Depression Not Otherwise Specified (NOS), or Dysthymia, as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV or DSM-V criteria
* Current depressive symptoms that warrant intervention as determined by a score of ≥ 11 on the Quick Inventory of Depressive Symptomatology - Clinician (QIDS-C)
* Able to communicate in spoken and written English
* Able and willing to provide written informed assent/consent and able to obtain written parental or guardian permission (if required, as specified in site standard operating procedure (SOP), by State law, and/or Institutional Review Board (IRB) policy) to be screened for and to enroll in IMPAACT 2002

Exclusion Criteria:

* Known or self-reported history of any psychotic disorder and/or bipolar I or II disorder
* Severe disorders (more than 6 symptoms) based on DSM-V criteria related to alcohol, cannabis or other substances; or those with moderate symptoms (4 or 5 symptoms) who are also currently experiencing withdrawal or dependence symptoms; within the past month prior to enrollment
* Per clinician assessment at screening, depression and/or suicidal ideation requiring more intensive treatment than the study provides or at immediate risk of being a danger to themselves or others
* Per participant report at screening, intends to relocate away from the study site during study participation
* Currently in therapy with a non-study provider, unless willing to switch to a study-trained provider
* Has any other condition that, in the opinion of the Investigator of Record (IoR)/designee, would preclude informed assent/consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Brown, MD, Study Chair — Rhode Island Hospital; Brown University
Locations (13):
- United States (13):
  - University of Southern California - MCA Center (CRS 5048),, Alhambra, California
  - University California, San Diego (CRS 4601), La Jolla, California
  - David Geffen School of Medicine at UCLA (CRS 5112), Los Angeles, California
  - Children's Hospital of Colorado (CRS 5052), Aurora, Colorado
  - Children's Diagnostic and Treatment Center (CRS 5055), Fort Lauderdale, Florida
  - Emory University School of Medicine (CRS 5030), Atlanta, Georgia
  - Rush University Medical Center (CRS 5083), Chicago, Illinois
  - Johns Hopkins University School of Medicine (CRS 5092), Baltimore, Maryland
  - Stony Brook University Medical Center (CRS 5040), Stony Brook, New York
  - Bronx-Lebanon Hospital Center (CRS 5114), The Bronx, New York
  - Jacobi Medical Center (CRS 5013), The Bronx, New York
  - St Jude Children's Research Hospital (CRS 6501), Memphis, Tennessee
  - Texas Children's/Baylor (CRS 3801), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data and related data dictionaries that underlie results in the publication will be shared after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT network,
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.
URL: https://www.impaactnetwork.org/studies/submit-research-proposal

REFERENCES:
- [Background] Brown LK, Kennard BD, Emslie GJ, Mayes TL, Whiteley LB, Bethel J, Xu J, Thornton S, Tanney MR, Hawkins LA, Garvie PA, Subramaniam GA, Worrell CJ, Stoff LW; Adolescent Trials Network for HIVAIDS Interventions. Effective Treatment of Depressive Disorders in Medical Clinics for Adolescents and Young Adults Living With HIV: A Controlled Trial. J Acquir Immune Defic Syndr. 2016 Jan 1;71(1):38-46. doi: 10.1097/QAI.0000000000000803. PMID 26761270
- [Background] Bernstein IH, Rush AJ, Trivedi MH, Hughes CW, Macleod L, Witte BP, Jain S, Mayes TL, Emslie GJ. Psychometric properties of the Quick Inventory of Depressive Symptomatology in adolescents. Int J Methods Psychiatr Res. 2010 Dec;19(4):185-94. doi: 10.1002/mpr.321. PMID 20683845
- See also: The Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (AE) (DAIDS AE Grading Table), Corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Richard M Selik, Eve D Mokotoff, Bernard Branson, et al. Revised Surveillance Case Definition for HIV Infection - United States, 2014. Morbidity and Mortality Weekly Report (MMWR) 2014; 63 (No. 3):7 — https://www.cdc.gov/mmwr/pdf/rr/rr6303.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS Expedited Adverse Events (EAE) Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Once enrollment opened (Dec 20, 2016), sites prepared lists of potential participants. The approach order was randomized in blocks of six. Sites were instructed to approach participants in order by block. A protocol letter of amendment in April 27, 2018 removed this requirement. First enrolled March 6, 2017, and the last enrolled on March 5, 2019
Pre-assignment Details: Sites were randomized to COMB-R or ESC with balancing based on information collected during application to participate and also in a pre-study survey, which gathered grouped data on characteristics of potential participants at each site including sex at birth, age group, mode of HIV transmission, HIV viral suppression status, level of depression.
Units Other Than Participants: sites
Period: Overall Study
Arm/Group | COMB-R | Enhanced Standard of Care
Started | 81; 6 sites (One additional site in the COMB-R group withdrew prior to the start of participant enrollment.) | 75; 7 sites
Week 24 Visit | 74; 6 sites (These are the numbers still on study at week 24) | 72; 7 sites
Completed (This is the completion information for the week 48 visit) | 70; 6 sites | 66; 7 sites
Not Completed | 11; 0 sites | 9; 0 sites
Not completed — Unable to get to clinic | 6 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — severe debilitation | 1 | 0
Not completed — Other | 0 | 1
Not completed — not willing to adhere to protocol | 2 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: site
Groups:
- Total: Total of all reporting groups
Arm/Group | COMB-R | Enhanced Standard of Care | Total
Number analyzed (Participants) | 81 | 75 | 156
Number analyzed (site) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (2.6) | 21.2 (3.0) | 21.4 (2.8)
Age, Customized [Count of Participants; unit: Participants]
  Age, categorized: 12-18 yrs | 14 | 19 | 33
  Age, categorized: 19-24 yrs | 67 | 56 | 123
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 38 | 82
  Male | 37 | 37 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, non-Hispanic | 5 | 3 | 8
  Race/Ethnicity: Black, Non- Hispanic | 51 | 38 | 89
  Race/Ethnicity: Hispanic, regardless of race | 19 | 33 | 52
  Race/Ethnicity: Asian, Pacific Islander | 2 | 0 | 2
  Race/Ethnicity: More than one race | 1 | 1 | 2
  Race/Ethnicity: Missing/Unknown | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81 | 75 | 156
Route of HIV acquisition [Count of Participants; unit: Participants]
  Perinatal | 40 | 43 | 83
  Behavioral | 41 | 32 | 73
log10 (HIV viral load copies/mL) [Mean (Standard Deviation); unit: log10 HIV copies/mL] | 2.2 (1.2) | 2.2 (1.3) | 2.2 (1.2)
QIDS-SR at study entry (mean) [Mean (Standard Deviation); unit: units on a scale] — QIDS-SR = Quick Inventory of Depression Symptomatology - Self Report. Scores range from 0 (least depression symptoms/severity) to 27 (highest level of depression symptoms/severity). Population: One participant had missing data or data which could not be scored
  units on a scale
    number analyzed (Participants) | 81 | 74 | 155
    (all) | 16.1 (4.1) | 13.8 (4.2) | 15 (4.3)
Taking psychiatric medications at study entry [Count of Participants; unit: Participants]
  not taking medications | 59 | 60 | 119
  taking psychiatric medications | 22 | 15 | 37
Average of site-level mean age [Mean (Standard Deviation); unit: years] — This measure is the average of the site-level mean ages within each treatment group.
  years | 21.5 (0.6) | 21.3 (1.8) | 21.4 (1.3)
Average of site-level % male [Mean (Standard Deviation); unit: percent] — This is the average of the site-level percent of male participants within each treatment group.
  percent | 44.9 (24.4) | 44.6 (24.5) | 44.7 (23.4)
Average of site-level % black participants [Mean (Standard Deviation); unit: percent] — This is the average of the site-level percents of Black participants within each treatment group.
  percent | 65.1 (40) | 57 (32.6) | 60.7 (34.9)
Average of site-level % with perinatal transmission [Mean (Standard Deviation); unit: percent] — This is the average of the site-level percentages of participants with perinatal HIV acquisition within treatment group.
  percent | 49.1 (26.3) | 56.2 (22.1) | 52.9 (23.4)
Average of site-level mean QIDS-SR scores [Mean (Standard Deviation); unit: units on a scale] — This measure is the average of the site-level mean QIDS-SR scores within treatment group. QIDS-SR = Quick Inventory of Depression Symptomatology - Self Report. Scores range from 0 (least depression symptoms/severity) to 27 (highest level of depression symptoms/severity).
  units on a scale | 16.2 (1.3) | 14.5 (3.2) | 15.3 (2.6)
Average of site-level mean log 10 (HIV viral load copies/mL) [Mean (Standard Deviation); unit: log10 HIV copies/mL] — This measure is the average of the site-level mean log10 HIV copes/mL within treatment group.
  log10 HIV copies/mL | 2.2 (0.7) | 2.1 (0.3) | 2.2 (0.5)
Average of site-level % of participants taking psychiatric medications [Mean (Standard Deviation); unit: percent] — This measure is the average of the site-level percentages of participants taking psychiatric medications within treatment group.
  percent | 28.0 (13.2) | 21.4 (19.0) | 24.5 (16.3)

OUTCOME MEASURES:

1. Primary Outcome: Depression Outcomes: Quick Inventory of Depression Symptomatology - Self Report (QIDS-SR) Score
Description: The QIDS-SR ranges from 0-27 and assesses the severity and number of depression symptoms. Data completed through the Audio Computer Assisted Interview (ACASI) system are used for this outcome. A lower score indicates fewer depression symptoms and lower depression symptom severity. Scores for all participants at a site were averaged. The site-specific averages were then analyzed.
Time Frame: Week 24
Population: All participants who entered QIDS-SR data into the ACASI system were analyzed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Groups:
- Enhanced Standard of Care: Enhanced Standard of Care (ESC)
  Ongoing psychopharmacological and psychosocial counseling and treatment for depression at HIV clinical treatment centers enhanced by providing clinicians with up-to-date information and didactic training
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 66 | 67
Number analyzed (site) | 6 | 7
units on a scale | 6.7 [3.7 to 9.7] | 10.6 [8.8 to 12.3]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Test type: Superiority — We tested the null hypothesis that the treatment group means were equal vs. not. The study was designed for at least 80% power to detect an effect size of 0.8 standard deviations (SD), which corresponded to a difference of four points. We assumed an intracluster correlation coefficient (ICC) between 0.02 and 0.16 and allowed for 10% non-evaluability. In a pre-planned interim analysis, we estimated the ICC based on the entry QIDS-SR to be 0.10; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = -3.86, 95% CI 2-sided [-6.79 to -0.94] — We subtracted the mean of the ESC group from the mean of the COMB-R group. Because a lower score indicated less severe depressive symptoms, a negative value indicated superiority

2. Primary Outcome: Depression Outcomes: Response to Treatment, Defined as a Decrease in QIDS-SR Score by >50%
Description: We are assessing the percentage of participants with a response to treatment.The percentage of participants at each site with a response was calculated. These percentages were averaged for each treatment and the treatment averages were compared. A response to treatment is considered a decrease in Quick Inventory of Depression Symptomatology, Self Report (QIDS-SR) from Study entry to Week 24 by more than 50%. The week 0 value is generally considered the entry value. Priority is given to the ACASI score at week 0. In certain cases, the week 1 ACASI value is used if there is no ACASI score at week 0, but there is one at week 1. Paper form scores are used for "study entry" if there is no ACASI record, with the value at week 0 prioritized over the value at week 1. Otherwise, ACASI data are used for this outcome. The QIDS-SR is scored from 0 to 27 with a lower score indicating less symptomatology.
Time Frame: Week 0 and Week 24
Population: We analyzed data from all participants with ACASI data at weeks 0 and 24.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 66 | 66
Number analyzed (site) | 6 | 7
percent | 62.3 [39 to 85.5] | 17.9 [7.0 to 28.9]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Test type: Superiority — We tested the null hypothesis that the treatment group means were equal vs. not; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 44.3, 95% CI 2-sided [23.1 to 65.5] — We subtracted the group mean of the site percents with response for the ESC group from that of the COMB-R group. A positive value indicates the COMB-R group had a higher mean percent of participants with response compared to the ESC group

3. Primary Outcome: Depression Outcomes: Remission, Defined as a QIDS-SR Score <= 5
Description: We computed the percentage of participants at each site with remission and then compared the percentages. Remission is defined as a Quick Inventory of Depression Symptomatology, self-report (QIDS-SR) score <= 5. ACASI data are used for this outcome. The QIDS-SR scale is from 0-27 with a lower score indicating tess symptomatology.
Time Frame: Week 24
Population: We analyzed data from all participants with an ACASI QIDS-SR score at week 24.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 66 | 67
Number analyzed (site) | 6 | 7
percent | 47.9 [22.7 to 73.0] | 17.0 [7.2 to 26.8]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Test type: Superiority — We tested the null hypothesis that the treatment group means were equal vs. not; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = 30.9, 95% CI 2-sided [8.9 to 52.9] — We subtracted the group mean of the site percents with remission for the ESC group from the COMB-R group so a positive value indicates the COMB-R group has more participants with remission

4. Primary Outcome: Biological Outcomes: Cluster of Differentiation 4 (CD4) Cell Count at Week 24
Description: CD4 cell counts are cells/microL (uL). CD4 cell counts of all participants at a site were averaged. The averages were then analyzed.
Time Frame: Week 24
Population: All participants with a CD4 cell count at week 24 were analyzed.
Measure: Mean (95% Confidence Interval); unit: cells/uL
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 66 | 71
Number analyzed (site) | 6 | 7
cells/uL | 703 [466 to 940] | 683 [524 to 842]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Test type: Superiority — We tested the null hypothesis that the treatment group means were equal vs. not; p = 0.86, t-test, 2 sided; Mean Difference (Final Values) = 19, 95% CI 2-sided [-223 to 262] — Group mean for ESC is subtracted from the group mean for COMB-R. The group means are the means of the site mean CD4 cell counts

5. Primary Outcome: Biological Outcomes: Plasma HIV RNA Level at Week 24
Description: Plasma HIV RNA data are calculated on the log10 scale as log10(RNA copies/mL)
  For this analysis, HIV-1 RNA values (copies per mL) that were censored below the lower limit of quantification (LLQ) were imputed to be equal to the LLQ - 1. The LLQ was considered to be 40 copies/mL. Viral load was calculated on the log10 scale as log10(RNA copies/mL). Viral load suppression was also measured as copies < 40.
  The log10 (RNA copies/mL) values were averaged by site and those averages were analyzed.
Time Frame: Week 24
Population: We analyzed data for all participants with a non-missing HIV RNA copies value at week 24.
Measure: Mean (95% Confidence Interval); unit: log10 HIV RNA (copies/mL)
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 67 | 73
Number analyzed (site) | 6 | 7
log10 HIV RNA (copies/mL) | 2.23 [1.48 to 2.97] | 2.06 [1.47 to 2.65]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Test type: Superiority — We tested the null hypothesis that the treatment group means were equal vs. not; p = 0.66, t-test, 2 sided; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.65 to 0.99] — We subtracted the group mean for the ESC group from the group mean of the COMB-R group. The group means are the means of the site mean log10 HIV RNA copies/mL

6. Secondary Outcome: Adherence Outcomes: Adherence to Anti-HIV Medications - Number of Days in Last 30 With Any Missed Doses
Description: Adherence to anti-HIV medications at each assessment for the first 24 weeks (during active treatment) and at 48 weeks, as measured by self-report. The first of three questions was to assess the number of days in the last 30 with any missed medication doses.The average number of days for all participants at a site were averaged. The site-specific averages were then analyzed.
Time Frame: Weeks 24 and 48
Population: We analyzed data for all participants with an ACASI interview at either week 24 or week 48
Measure: Mean (95% Confidence Interval); unit: days
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 60 | 65
Number analyzed (site) | 6 | 7
days
  week 24 | 4.4 [2.6 to 6.2] | 2.3 [1.0 to 3.7]
  week 48: number analyzed (Participants) | 58 | 60
  week 48 | 4.8 [1.1 to 8.5] | 4.7 [0.4 to 9.0]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, number of days in last 30 with any missed HIV medication doses reported at week 24; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [0.1 to 4.0] — A positive difference indicates COMB-R group had a site-level average of more days in last 30 with missed HIV medication doses
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, number of days in last 30 with any missed HIV medication doses reported at week 48; Test type: Superiority; p = 0.96, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-5.0 to 5.2] — A positive difference reflects greater number of days with missed HIV medication doses in last 30 days for COMB-R group

7. Secondary Outcome: Adherence Outcomes: Adherence to Anti-HIV Medications - How Good Participant Was at Taking Medicines as Instructed
Description: Adherence to anti-HIV medications at each assessment for the first 24 weeks (during active treatment) and at 48 weeks, as measured by self-report. The second of three questions was how good the participant is at taking his medication as instructed in the last 30 days. Response scales are Likert from 1 to 6, with a higher score indicating better adherence. 1=Very poor .... 6=Excellent. The average score for all participants at each site was computed and these site-level summaries were compared across treatments.
Time Frame: Weeks 24 and 48
Population: We analyzed data for each participants with a response at either week 24 or week 48.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 63 | 69
Number analyzed (site) | 6 | 7
units on a scale
  Week 24 | 4.3 [3.8 to 4.9] | 4.7 [4.1 to 5.4]
  Week 48: number analyzed (Participants) | 59 | 63
  Week 48 | 4.4 [3.7 to 5.1] | 4.2 [3.9 to 4.5]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, how good was participant at taking HIV medication doses; reported at week 24; Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.4] — A positive difference means the COMB-R group rated adherence to HIV medications better than the ESC group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, how good was participant at taking HIV medication doses; reported at week 48; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.9] — A positive difference would indicate the COMB-R group rated their adherence better than the ESC group

8. Secondary Outcome: Adherence Outcomes: Adherence to Anti-HIV Medications - How Often Did Participant Take Medications as Instructed
Description: Adherence to anti-HIV medications at each assessment for the first 24 weeks (during active treatment) and at 48 weeks, as measured by self-report. The third of three questions was how often the participant took medication correctly in the last 30 days. Response scales are Likert from 1 to 6, with a higher score indicating better adherence. 1=Never ... 6=Always. The average score for all participants at a site was computed and these site-level summaries were compared across treatments.
Time Frame: Weeks 24 and 48
Population: We analyzed data for all participants with adherence reported at either week 24 or week 48
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 62 | 69
Number analyzed (site) | 6 | 7
units on a scale
  Week 24 | 4.8 [4.3 to 5.3] | 5.2 [4.7 to 5.7]
  Week 48: number analyzed (Participants) | 59 | 63
  Week 48 | 4.8 [3.9 to 5.6] | 4.5 [3.9 to 5.1]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, how often did participant take HIV medication as instructed; reported at week 24; Test type: Superiority; p = 0.14, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.1 to 0.2] — A positive difference would indicate the COMB-R group rated their adherence better than the ESC group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, how often did participant take HIV medication as instructed; reported at week 48; Test type: Superiority; p = 0.49, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.6 to 1.1] — A positive difference would indicate the COMB-R group rated their adherence better than the ESC group

9. Secondary Outcome: Adherence Outcomes: Adherence to Psychiatric Medications - Number of Days in Last 30 With Any Missed Doses
Description: Adherence to depression medications at each assessment for the first 24 weeks (during active treatment) and at 48 weeks, as measured by self-report for those participants taking depression medications. Three questions were asked; The first of the three questions was to assess the number of days in the last 30 with any missed medication doses.The average number of days for all participants at a site were averaged. The site-specific averages were then analyzed.
Time Frame: Weeks 24 and 48
Population: We analyzed data for all participants with adherence to depression medication data reported at either week 24 or week 48. Participants not taking depression medication were excluded.
Measure: Mean (95% Confidence Interval); unit: days
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 28 | 21
Number analyzed (site) | 6 | 7
days
  week 24: number analyzed (Participants) | 28 | 18
  week 24 | 3.4 [0.9 to 5.9] | 1.2 [0.1 to 2.2]
  week 48: number analyzed (Participants) | 20 | 21
  week 48 | 3.6 [1.1 to 6.2] | 6.4 [-3.4 to 16.1]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, number of days in last 30 with any missed depression medication doses reported at week 24; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [0.0 to 4.4] — A positive difference would indicate those in the COMB-R group had more days with missed depression medications than those in the ESC group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, number of days in last 30 with any missed depression medication doses reported at week 48; Test type: Superiority; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-12.5 to 7.1] — A positive difference would indicate those in the COMB-R group reported more days with missed doses than those in the ESC group

10. Secondary Outcome: Adherence Outcomes: Adherence to Psychiatric Medications - How Good Participant Was at Taking Medications as Instructed
Description: Adherence to depression medications at each assessment for the first 24 weeks (during active treatment) and at 48 weeks, as measured by self-report tor those participants taking depression medications. The second of three questions was how good the participant is at taking his medication as instructed during the last 30 days. Response scales are Likert from 1 to 6, with a higher score indicating better adherence.1=Very poor .... 6=Excellent. The average score for all participants at each site was computed and these site-level summaries were compared across treatments.
Time Frame: Weeks 24 and 48
Population: We analyzed data for all participants with adherence to depression medications reported at either week 24 or week 48. Participants not on depression medications were excluded.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 27 | 21
Number analyzed (site) | 6 | 7
units on a scale
  week 24: number analyzed (Participants) | 27 | 18
  week 24 | 4.5 [4.0 to 5.1] | 5.2 [4.4 to 5.9]
  week 48: number analyzed (Participants) | 20 | 21
  week 48 | 4.5 [3.8 to 5.2] | 4.0 [2.6 to 5.5]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, how good was participant at taking depression medication; reported at week 24; Test type: Superiority; p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.5 to 0.2] — A positive difference would indicate those in the COMB-R group were better at taking medications
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, how good was participant at taking depression medication; reported at week 48; Test type: Superiority; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.1 to 2.0] — A positive difference would indicate those in the COMB-R group were better at taking their medications

11. Secondary Outcome: Adherence Outcomes: Adherence to Psychiatric Medications - How Often Did Participant Take Medicines as Instructed
Description: Adherence to depression medications at each assessment for the first 24 weeks (during active treatment) and at 48 weeks, as measured by self-report for those participants taking depression medications. The third of three questions was how often the participant took medication correctly in the past 30 days. Response scales are Likert from 1 to 6, with a higher score indicating better adherence: 1=Never .... 6=Always. The average score for all participants at each site was computed and these site-level summaries were compared across treatments.
Time Frame: Weeks 24 and 48
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 27 | 21
Number analyzed (site) | 6 | 7
units on a scale
  Week 24: number analyzed (Participants) | 27 | 18
  Week 24 | 4.8 [4.1 to 5.5] | 5.4 [5.0 to 5.8]
  Week 48: number analyzed (Participants) | 20 | 21
  Week 48 | 5.1 [4.5 to 5.6] | 4.3 [2.7 to 5.9]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, how often did participant take depression medication as instructed; reported at week 24; Test type: Superiority; p = 0.07, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.3 to 0.1] — A positive difference would indicate those in the COMB-R group reported better adherence
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; Comparison of COMB-R and ESC groups, how often did participant take depression medication as instructed; reported at week 48; Test type: Superiority; p = 0.28, t-test, 2 sided; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-0.8 to 2.3] — A positive difference would indicate those in the COMB-R group reported better adherence than those in the ESC group

12. Secondary Outcome: Adherence Outcomes: Adherence to Psychotherapy Sessions
Description: We computed the number of scheduled counseling sessions attended. The average number of sessions was computed for all participants at each site and these site-level averages were compared across treatments.Where study visits for weeks 0 and 1 were held on the same day, the counseling session for week 1 would have been administered at week 0.
Time Frame: Weeks 1, 6, 12 and 24
Population: We analyzed the number of sessions for all participants entering the study.
Measure: Mean (95% Confidence Interval); unit: sessions
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 81 | 75
Number analyzed (site) | 6 | 7
sessions | 3.5 [3.3 to 3.8] | 3.7 [3.3 to 4.0]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.3]

13. Secondary Outcome: Adherence Outcomes: Adherence to COMB-R Medication Management Sessions
Description: We computed the number of scheduled medication management sessions (COMB-R only) attended. The average number of sessions was computed for all participants at each site. We took the mean of the site-level averages.
Time Frame: Weeks 1, 6, 12 and 24
Population: We analyzed data for all COMB-R participants.
Measure: Mean (Standard Deviation); unit: sessions
Units Other Than Participants: site
Arm/Group | COMB-R
Number analyzed (Participants) | 81
Number analyzed (site) | 6
sessions | 3.6 (0.2)

14. Secondary Outcome: Adherence Outcomes: Adherence to Study Visits
Description: We computed the number study visits completed as the number of scheduled study visits completed to date as of week 24 and week 48. However in some cases, weeks 0 and 1 visits were done on the same day. In that case, they were counted as separate visits.The average number of visits was computed for all participants at each site and these site-level averages were compared across treatments.
Time Frame: Weeks 0, 1, 6, 12, 24, 36 and 48
Population: We analyzed data for all study participants
Measure: Mean (95% Confidence Interval); unit: visits
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 81 | 75
Number analyzed (site) | 6 | 7
visits
  week 24 | 4.7 [4.5 to 4.9] | 4.7 [4.4 to 5.1]
  week 48 | 6.4 [6.0 to 6.8] | 6.5 [6.0 to 7.0]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The average number of scheduled study visits through week 24 was computed for each site. The analysis was of these site-level averages. These values were compared between study groups; Test type: Superiority; p = 0.67, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; We computed the average number of scheduled study visits through week 48 for each site. We then averaged the site-level values and compared study groups; Test type: Superiority; p = 0.74, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.5]

15. Secondary Outcome: Depression Outcomes: Quick Inventory of Depression Symptomatology Self-Report (QIDS-SR) Score Over 48 Weeks.
Description: The Quick Inventory of Depression Symptomatology Self-Report (QIDS-SR) score ranges from 0-27 and assesses the severity and number of depression symptoms. Data completed through the Audio Computer Assisted Interview (ACASI) system were used for this outcome. A lower score indicates fewer depression symptoms and lower depression symptom severity. Scores for all participants at a site were averaged. The site-specific averages were then analyzed.
Time Frame: Week 48
Population: We analyzed all data from participants with a QIDS-SR score at week 48.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 68 | 59
Number analyzed (site) | 6 | 7
units on a scale | 7.09 [5.05 to 9.13] | 9.08 [6.79 to 11.36]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; We tested the null hypothesis that the treatment group means were equal vs. not; Test type: Superiority; p = 0.14, t-test, 2 sided; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-4.74 to 0.76] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Depression Outcomes: Quick Inventory of Depression Symptomatology Self-Report (QIDS-SR) Response to Treatment Over 48 Weeks, Defined as a Decrease in QIDS-SR Score by > 50%
Description: A response to treatment was considered to be a decrease in Quick Inventory of Depression Symptomatology, Self Report (QIDS-SR) from Study entry to Week 48 by more than 50%. The week 0 value was generally considered the entry value. Priority was given to the ACASI score at week 0. In certain cases, the week 1 ACASI value was used if there was no ACASI score at week 0, but there was one at week 1. Paper form scores were used for "study entry" if there were no ACASI records, with the value at week 0 prioritized over the value at week 1. Otherwise, ACASI data were used for this outcome. The QIDS-SR was scored from 0 to 27 with a lower score indicating less symptomatology.The percentage of participants with a QIDS-SR response at each site was calculated. These percentages were averaged for each treatment and the treatment averages were compared.
Time Frame: Week 0 and Week 48
Population: We analyzed data from participants with ACASI data at weeks 0 and 48.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 68 | 58
Number analyzed (site) | 6 | 7
percent | 58.7 [38.7 to 78.7] | 33.4 [13.8 to 53.0]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; We tested the null hypothesis that the treatment group means were equal vs. not; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 25.3, 95% CI 2-sided [0.5 to 50.0] — [estimate comment as in outcome 2, analysis 1]

17. Secondary Outcome: Depression Outcomes: Quick Inventory of Depression Symptomatology Self-Report (QIDS-SR) Score Remission Over 48 Weeks
Description: Remission is defined as a Quick Inventory of Depression Symptomatology, self-report (QIDS-SR) score of 5 or less. ACASI data are used for this outcome. The QIDS-SR scale is from 0-27 with a lower score indicating tower depression symptomatology. We computed the percentage of participants at each site with remission and then compared the site-level percentages across treatments.
Time Frame: Week 48
Population: We analyzed data for all participants with a week 48 QIDS-SR ACASI score.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 68 | 59
Number analyzed (site) | 6 | 7
percent | 43.7 [20.3 to 67.1] | 27.5 [5.2 to 49.8]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; We tested the null hypothesis that the treatment group means were equal vs. not; Test type: Superiority; p = 0.24, t-test, 2 sided; Mean Difference (Final Values) = 16.3, 95% CI 2-sided [-12.3 to 44.8] — [estimate comment as in outcome 3, analysis 1]

18. Secondary Outcome: Effect of Demographic, Behavioral, and Biological Modifiers on Depression Outcomes: Quick Inventory of Depression Symptomatology (QIDS-SR) Score
Description: QIDS-SR score (defined in Outcome 15). Effect of moderators on depression outcomes:Demographic: age group, gender, mode of HIV acquisition, initial level of depression (QIDS-SR categorized as severe/very severe vs. moderate or less severity); Biological: baseline CD4 (count/uL categorized as stage 3 [< 200 cells] vs. less than stage 3), nadir CD4 at study entry (based on count/uL and considering worst classification across ages, defined below), plasma HIV RNA suppression status, Center for Disease Control and Prevention (CDC) clinical stage at entry (Stage 3 vs. less than stage 3): Determination of nadir CD4 cell count as Stage 3 was based on the following: If any of the following were true, the overall CD4 nadir cell count was classified as Stage 3: <750 cells at < 1 year of age; < 500 cells at 1-5 years of age; <200 cells at 6+ years of age (from Revised Surveillance Case Definition for HIV Infection - United States, 2014). See analysis section for description of method.
Time Frame: Week 48
Population: All participants in each effect modifier subgroup with ACASI data at week 48 were analyzed. In some cases a site did not have any participants in a given subgroup, in which case an interaction term for that site could not be computed and the site was excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 68 | 59
Number analyzed (site) | 6 | 7
units on a scale
  Sex at birth - Male: number analyzed (Participants) | 32 | 28
  Sex at birth - Male: number analyzed (site) | 6 | 6
  Sex at birth - Male | 8.15 [3.19 to 13.11] | 6.11 [3.34 to 8.89]
  Sex at birth- Female: number analyzed (Participants) | 36 | 31
  Sex at birth- Female | 6.78 [3.88 to 9.67] | 11.53 [8.81 to 14.24]
  Age group - Younger (12-18 years): number analyzed (Participants) | 14 | 13
  Age group - Younger (12-18 years): number analyzed (site) | 6 | 6
  Age group - Younger (12-18 years) | 6.57 [4.60 to 8.53] | 10.13 [4.94 to 15.31]
  Age Group - Older (19-24 years): number analyzed (Participants) | 54 | 46
  Age Group - Older (19-24 years) | 7.00 [4.38 to 9.62] | 8.50 [5.81 to 11.18]
  Viral Suppression - Suppressed (less than 40 copies/mL): number analyzed (Participants) | 41 | 31
  Viral Suppression - Suppressed (less than 40 copies/mL) | 5.88 [3.01 to 8.75] | 9.80 [6.13 to 13.46]
  Viral Suppression - Not Suppressed (40 copies/mL or more): number analyzed (Participants) | 27 | 28
  Viral Suppression - Not Suppressed (40 copies/mL or more) | 7.06 [3.13 to 10.98] | 8.21 [5.80 to 10.62]
  QIDS-SR - Severe/Very severe: number analyzed (Participants) | 40 | 19
  QIDS-SR - Severe/Very severe: number analyzed (site) | 6 | 6
  QIDS-SR - Severe/Very severe | 8.51 [6.24 to 10.79] | 11.19 [6.06 to 16.31]
  QIDS-SR - Mild/Moderate: number analyzed (Participants) | 28 | 39
  QIDS-SR - Mild/Moderate: number analyzed (site) | 6 | 6
  QIDS-SR - Mild/Moderate | 5.46 [3.34 to 7.57] | 7.94 [6.07 to 9.82]
  Transmission - Perinatal: number analyzed (Participants) | 32 | 33
  Transmission - Perinatal | 7.61 [5.73 to 9.48] | 9.81 [6.13 to 13.50]
  Transmission- Behavioral: number analyzed (Participants) | 36 | 26
  Transmission- Behavioral | 7.31 [3.90 to 10.72] | 9.21 [5.34 to 13.08]
  CDC Stage 3: number analyzed (Participants) | 12 | 13
  CDC Stage 3: number analyzed (site) | 4 | 5
  CDC Stage 3 | 8.25 [3.68 to 12.82] | 6.22 [3.37 to 9.06]
  CDC Less than Stage 3: number analyzed (Participants) | 56 | 46
  CDC Less than Stage 3 | 7.63 [4.40 to 10.86] | 9.18 [6.86 to 11.51]
  CD4 Stage 3 (less than 200 cells/uL): number analyzed (Participants) | 6 | 6
  CD4 Stage 3 (less than 200 cells/uL): number analyzed (site) | 3 | 3
  CD4 Stage 3 (less than 200 cells/uL) | 10.00 [-0.83 to 20.83] | 5.56 [-1.87 to 12.98]
  CD4 - Less than Stage 3 (200 cells/uL or more): number analyzed (Participants) | 62 | 52
  CD4 - Less than Stage 3 (200 cells/uL or more) | 6.66 [4.98 to 8.35] | 9.14 [7.10 to 11.18]
  CD4 Nadir Stage 3: number analyzed (Participants) | 19 | 18
  CD4 Nadir Stage 3: number analyzed (site) | 6 | 5
  CD4 Nadir Stage 3 | 6.05 [2.85 to 9.24] | 9.18 [3.23 to 15.13]
  CD4 Nadir - Less than Stage 3: number analyzed (Participants) | 49 | 41
  CD4 Nadir - Less than Stage 3 | 7.68 [4.31 to 11.05] | 9.24 [7.37 to 11.12]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; An interaction effect is computed based on subgroup differences within sites. The mean subgroup difference is computed for each treatment group and the interaction effect is the difference of those group mean differences. This is equivalent to taking the differences of the treatment effects between subgroups. Note: For QIDS-SR, since a lower score reflects fewer depression symptoms, a positive treatment effect is a negative difference value between groups; Test type: Superiority; p = 0.01, t-test, 2 sided — This is the test of effect modification by sex at birth; Mean Difference (Final Values) = 6.79, 95% CI 2-sided [2.30 to 11.28] — A positive value indicates that the treatment difference (lower QIDS-SR score with COMB-R than with ESC) was greater for females compared to males
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; An interaction effect is computed based on subgroup differences within sites. The mean subgroup difference is computed for each treatment group and the interaction effect is the difference of those group mean differences.This is equivalent to taking the differences of the treatment effects between subgroups. Note: For QIDS-SR, since a lower score reflects fewer depression symptoms, a positive treatment effect is a negative difference value between groups; Test type: Superiority; p = 0.23, t-test, 2 sided — This is the test of effect modification by age group; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-7.05 to 1.93] — A negative value indicates the treatment difference is greater for younger compared to older participants
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; An interaction effect is computed based on subgroup differences within sites. The mean subgroup difference is computed for each treatment group and the interaction effect is the difference of those group mean differences.This is equivalent to taking the differences of the treatment effects between subgroups.Note: For QIDS-SR, since a lower score reflects fewer depression symptoms, a positive treatment effect is a negative difference value between groups; Test type: Superiority; p = 0.31, t-test, 2 sided — This is the test of the effect modification of viral suppression status; Mean Difference (Final Values) = -2.77, 95% CI 2-sided [-8.48 to 2.95] — A negative value indicates a greater treatment difference among those with viral suppression at study entry compared to those without viral suppression
Statistical Analysis 4: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 18, analysis 3]; Test type: Superiority; p = 0.72, t-test, 2 sided — This is the test of effect modification by QIDS-SR depression level at study entry; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-4.29 to 5.95] — A positive value indicates a greater treatment difference among those with moderate levels of depression compared to severe depression
Statistical Analysis 5: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 18, analysis 2]; Test type: Superiority; p = 0.91, t-test, 2 sided — This is the test of effect modification by mode of transmission; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-5.91 to 5.31] — A negative value would indicate a greater treatment difference for those with perinatal HIV acquisition compared to behavioral acquisition
Statistical Analysis 6: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 18, analysis 2]; Test type: Superiority; p = 0.57, t-test, 2 sided — This is the test of effect modification by HIV CDC stage level; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [-3.91 to 6.57] — A positive value would indicate a greater treatment effect for those with less than HIV CDC Stage 3 compared to those with CDC Stage 3 HIV illness
Statistical Analysis 7: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 18, analysis 2]; Test type: Superiority; p = 0.10, t-test, 2 sided — This is the test of effect modification of CD4 Stage 3 at entry; Mean Difference (Final Values) = 5.93, 95% CI 2-sided [-1.73 to 13.59] — A positive value indicates a greater treatment effect among those with less than Stage 3 CD4 count at entry compared to those with Stage 3 CD4 count
Statistical Analysis 8: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 18, analysis 2]; Test type: Superiority; p = 0.58, t-test, 2 sided — This is the test of effect modification by Nadir Stage 3 level at study entry; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-7.74 to 4.60] — A negative value indicates a greater treatment effect among those with Stage 3 Nadir CD4 compare to those with less than Stage 3 Nadir CD4

19. Secondary Outcome: Effect of Demographic, Behavioral, and Biological Modifiers on Depression Outcomes: Response to Treatment
Description: Response to Treatment (defined in Outcome 16): Effect of moderators on depression outcomes: Demographic: age group, gender, mode of HIV acquisition, initial level of depression (QIDS-SR categorized as severe/very severe vs. moderate or less severity); Biological: baseline CD4 (count/uL categorized as stage 3 [< 200 cells] vs. less than stage 3), nadir CD4 at study entry (based on count/uL and considering worst classification across ages, defined below), plasma HIV RNA suppression status, Center for Disease Control and Prevention (CDC) clinical stage at entry (Stage 3 vs. less than stage 3): Determination of nadir CD4 cell count as Stage 3 was based on the following: If any of the following were true, the overall CD4 nadir cell count was classified as Stage 3: <750 cells at < 1 year of age; < 500 cells at 1-5 years of age; <200 cells at 6+ years of age (from Revised Surveillance Case Definition for HIV Infection - United States, 2014). See analysis section for description of method.
Time Frame: Week 0 and Week 48
Population: We analyzed data for every participant with a defined response. In order to have a defined QIDS-SR response the participant had to have data at both week 0 and week 48. In some cases a site did not have any participants in a given subgroup, in which case an interaction term for that site could not be computed and the site was excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 68 | 58
Number analyzed (site) | 6 | 7
percent
  Sex at birth- Male: number analyzed (Participants) | 32 | 28
  Sex at birth- Male: number analyzed (site) | 6 | 6
  Sex at birth- Male | 54.95 [14.40 to 95.51] | 67.30 [33.24 to 101.36]
  Sex at birth - Female: number analyzed (Participants) | 36 | 30
  Sex at birth - Female | 64.58 [35.12 to 94.05] | 7.82 [-1.60 to 17.24]
  Age group - Younger (12-18 years): number analyzed (Participants) | 14 | 13
  Age group - Younger (12-18 years): number analyzed (site) | 6 | 6
  Age group - Younger (12-18 years) | 71.11 [29.92 to 112.30] | 22.22 [-4.11 to 48.56]
  Age group - Older (19-24 years): number analyzed (Participants) | 54 | 45
  Age group - Older (19-24 years) | 56.28 [33.16 to 79.39] | 43.25 [13.37 to 73.13]
  Viral status - Suppressed (less than 40 copies /mL): number analyzed (Participants) | 41 | 31
  Viral status - Suppressed (less than 40 copies /mL) | 66.61 [38.97 to 94.26] | 37.93 [11.41 to 64.44]
  Viral status - Not Suppressed (40 or more copies/mL): number analyzed (Participants) | 27 | 27
  Viral status - Not Suppressed (40 or more copies/mL): number analyzed (site) | 6 | 6
  Viral status - Not Suppressed (40 or more copies/mL) | 55.46 [25.21 to 85.71] | 35.28 [-0.40 to 70.96]
  Depression status - Severe/very severe: number analyzed (Participants) | 40 | 19
  Depression status - Severe/very severe: number analyzed (site) | 6 | 6
  Depression status - Severe/very severe | 55.45 [28.50 to 82.39] | 30.56 [-11.45 to 72.56]
  Depression status- Mild/Moderate: number analyzed (Participants) | 28 | 39
  Depression status- Mild/Moderate: number analyzed (site) | 6 | 6
  Depression status- Mild/Moderate | 58.33 [36.91 to 79.75] | 41.31 [27.67 to 54.96]
  Mode of transmission - Perinatal: number analyzed (Participants) | 32 | 32
  Mode of transmission - Perinatal: number analyzed (site) | 6 | 6
  Mode of transmission - Perinatal | 57.14 [33.41 to 80.88] | 15.00 [-9.61 to 39.61]
  Mode of transmission - Behavioral: number analyzed (Participants) | 36 | 26
  Mode of transmission - Behavioral | 57.44 [21.50 to 93.38] | 48.81 [7.74 to 89.88]
  CDC Stage 3: number analyzed (Participants) | 12 | 13
  CDC Stage 3: number analyzed (site) | 4 | 5
  CDC Stage 3 | 78.13 [37.12 to 119.13] | 50.00 [3.73 to 96.27]
  CDC less than Stage 3: number analyzed (Participants) | 56 | 45
  CDC less than Stage 3 | 48.52 [15.68 to 81.36] | 40.63 [10.86 to 70.41]
  CD4 Stage 3 (less than 200 cells/uL): number analyzed (Participants) | 6 | 6
  CD4 Stage 3 (less than 200 cells/uL): number analyzed (site) | 3 | 3
  CD4 Stage 3 (less than 200 cells/uL) | 61.11 [-25.07 to 147.30] | 38.89 [-47.30 to 125.07]
  CD4 - less than stage 3 (200 or more cells/uL): number analyzed (Participants) | 62 | 51
  CD4 - less than stage 3 (200 or more cells/uL) | 59.10 [39.48 to 78.73] | 34.85 [15.03 to 54.68]
  Nadir CD4 Stage 3: number analyzed (Participants) | 19 | 18
  Nadir CD4 Stage 3: number analyzed (site) | 6 | 5
  Nadir CD4 Stage 3 | 86.31 [61.63 to 110.99] | 23.00 [-5.31 to 51.31]
  Nadir CD4 - less than Stage 3: number analyzed (Participants) | 49 | 40
  Nadir CD4 - less than Stage 3 | 50.79 [24.09 to 77.49] | 37.11 [16.69 to 57.54]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; An interaction effect is computed based on subgroup differences within sites. The mean subgroup difference is computed for each treatment group and the interaction effect is the difference of those group mean differences. This is equivalent to taking the differences of the treatment effects between subgroups. Note: For the percent of participants with QIDS-SR response, a positive treatment effect is a positive difference between groups; Test type: Superiority; p = 0.01, t-test, 2 sided — This is the test of effect modification by sex at birth; Mean Difference (Final Values) = -67.81, 95% CI 2-sided [-116.53 to -19.10] — A negative value indicates a greater treatment response (higher percent with response in COMB-R than in ESC group) among females compared to males
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.09, t-test, 2 sided — This is the test of effect modification by age group; Mean Difference (Final Values) = 43.08, 95% CI 2-sided [-8.23 to 94.38] — A positive value reflects a greater treatment effect among younger participants compared to older participants
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.93, t-test, 2 sided — This is the test of effect modification by viral suppression status; Mean Difference (Final Values) = 2.18, 95% CI 2-sided [-51.13 to 55.49] — A positive value would reflect a greater treatment response among those with suppressed viral status at entry compared to those without viral suppression
Statistical Analysis 4: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.87, t-test, 2 sided — This is the test of effect modification by entry QIDS-SR depression level; Mean Difference (Final Values) = 3.36, 95% CI 2-sided [-42.28 to 49.00] — A positive value would indicate a greater treatment response for those with severe depressive symptoms at study entry compared to those with moderate depression
Statistical Analysis 5: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.17, t-test, 2 sided — This is the test of effect modification by mode of transmission; Mean Difference (Final Values) = 41.65, 95% CI 2-sided [-21.91 to 105.20] — A positive value would indicate a larger treatment response for those with perinatal transmission compared to behavioral
Statistical Analysis 6: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.17, t-test, 2 sided — This is the test of effect modification by HIV CDC stage; Mean Difference (Final Values) = 49.40, 95% CI 2-sided [-26.02 to 124.83] — A positive value reflects a greater treatment response for those with HIV CDC Stage 3 classification compared to those with CDC classification less than Stage 3
Statistical Analysis 7: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.71, t-test, 2 sided — This is the test of effect modification by CD4 Stage at study entry; Mean Difference (Final Values) = 11.69, 95% CI 2-sided [-70.76 to 94.15] — A positive value would reflect greater treatment response for those with CD4 Stage 3 compared to those with less than Stage 3 CD4
Statistical Analysis 8: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.02, t-test, 2 sided — This is the test of effect modification by CD4 Nadir stage at study entry; Mean Difference (Final Values) = 52.48, 95% CI 2-sided [10.46 to 94.50] — A positive value reflects a larger treatment response among those with Stage 3 Nadir CD4 compared to those with less than Stage 3 Nadir CD4

20. Secondary Outcome: Effect of Demographic, Behavioral, and Biological Modifiers on Depression Outcomes: Remission
Description: Remission (defined in Outcome 17): Effect of moderators on depression outcomes: Demographic: age group, gender, mode of HIV acquisition, initial level of depression (QIDS-SR categorized as severe/very severe vs. moderate or less severity); Biological: baseline CD4 (count/uL categorized as stage 3 [< 200 cells] vs. less than stage 3), nadir CD4 at study entry (based on count/uL and considering worst classification across ages, defined below), plasma HIV RNA suppression status, Center for Disease Control and Prevention (CDC) clinical stage at entry (Stage 3 vs. less than stage 3): Determination of nadir CD4 cell count as Stage 3 was based on the following: If any of the following were true, the overall CD4 nadir cell count was classified as Stage 3: <750 cells at < 1 year of age; < 500 cells at 1-5 years of age; <200 cells at 6+ years of age (from Revised Surveillance Case Definition for HIV Infection - United States, 2014). See analysis section for description of method.
Time Frame: Week 48
Population: We analyzed data for all participants with an ACASI QIDS-SR reported at week 48. We computed the percent of participants with remission at week 48 at each site. In some cases a site did not have any participants in a given subgroup, in which case an interaction term for that site could not be computed and the site was excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 68 | 59
Number analyzed (site) | 6 | 7
percent
  Sex at Birth- Male: number analyzed (Participants) | 32 | 28
  Sex at Birth- Male: number analyzed (site) | 6 | 6
  Sex at Birth- Male | 44.54 [14.29 to 74.79] | 56.59 [11.32 to 101.85]
  Sex at birth - Female: number analyzed (Participants) | 36 | 31
  Sex at birth - Female | 42.13 [5.61 to 78.65] | 7.82 [-1.60 to 17.24]
  Age Group - Younger (12-18 years): number analyzed (Participants) | 14 | 13
  Age Group - Younger (12-18 years): number analyzed (site) | 6 | 6
  Age Group - Younger (12-18 years) | 31.11 [-7.63 to 69.85] | 22.22 [-4.11 to 48.56]
  Age Group - Older (19-24 years): number analyzed (Participants) | 54 | 46
  Age Group - Older (19-24 years) | 47.94 [20.03 to 75.86] | 34.68 [1.90 to 67.47]
  Viral Suppression - Suppressed (less than 40 copies/mL): number analyzed (Participants) | 41 | 31
  Viral Suppression - Suppressed (less than 40 copies/mL) | 49.84 [18.21 to 81.47] | 28.74 [1.28 to 56.20]
  Viral Suppression - not suppressed ( 40 copies/mL or more): number analyzed (Participants) | 27 | 28
  Viral Suppression - not suppressed ( 40 copies/mL or more) | 45.74 [2.93 to 88.55] | 30.24 [-1.00 to 61.48]
  QIDS-SR level - Severe/Very severe: number analyzed (Participants) | 40 | 19
  QIDS-SR level - Severe/Very severe: number analyzed (site) | 6 | 6
  QIDS-SR level - Severe/Very severe | 32.79 [8.18 to 57.41] | 27.78 [-14.59 to 70.14]
  QIDS-SR level - Mild/Moderate: number analyzed (Participants) | 28 | 39
  QIDS-SR level - Mild/Moderate: number analyzed (site) | 6 | 6
  QIDS-SR level - Mild/Moderate | 58.33 [36.91 to 79.75] | 35.76 [13.23 to 58.28]
  Mode of transmission - Perinatal: number analyzed (Participants) | 32 | 33
  Mode of transmission - Perinatal | 35.32 [13.03 to 57.61] | 16.43 [-3.68 to 36.53]
  Mode of transmission - Behavioral: number analyzed (Participants) | 36 | 26
  Mode of transmission - Behavioral | 39.85 [4.84 to 74.85] | 30.95 [-5.46 to 67.36]
  CDC Stage 3: number analyzed (Participants) | 12 | 13
  CDC Stage 3: number analyzed (site) | 4 | 5
  CDC Stage 3 | 40.63 [-37.89 to 119.14] | 56.67 [11.33 to 102.01]
  Less than CDC Stage 3: number analyzed (Participants) | 56 | 46
  Less than CDC Stage 3 | 36.30 [7.43 to 65.16] | 23.17 [4.17 to 42.18]
  CD4 Stage 3 (less than 200 cells/uL): number analyzed (Participants) | 6 | 6
  CD4 Stage 3 (less than 200 cells/uL): number analyzed (site) | 3 | 3
  CD4 Stage 3 (less than 200 cells/uL) | 44.44 [-82.04 to 170.93] | 55.56 [-70.93 to 182.04]
  CD4- less than Stage 3 (200 or more cells/uL): number analyzed (Participants) | 62 | 52
  CD4- less than Stage 3 (200 or more cells/uL) | 45.67 [22.58 to 68.76] | 24.85 [3.37 to 46.33]
  CD4 Nadir Stage 3: number analyzed (Participants) | 19 | 18
  CD4 Nadir Stage 3: number analyzed (site) | 6 | 5
  CD4 Nadir Stage 3 | 50.60 [1.19 to 100.00] | 28.00 [-4.14 to 60.14]
  CD4 Nadir- less than Stage 3: number analyzed (Participants) | 49 | 41
  CD4 Nadir- less than Stage 3 | 38.03 [9.61 to 66.45] | 26.40 [4.66 to 48.14]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; An interaction effect is computed based on subgroup differences within sites. The mean subgroup difference is computed for each treatment group and the interaction effect is the difference of those group mean differences. This is equivalent to taking the differences of the treatment effects between subgroups. Note: For the percent of participants with QIDS-SR remission, a positive treatment effect is a positive difference between groups; Test type: Superiority; p = 0.09, t-test, 2 sided — This is the test of effect modification by sex at birth; Mean Difference (Final Values) = -45.06, 95% CI 2-sided [-97.84 to 7.72] — A negative value indicates a greater treatment effect (higher percent with remission for COMB-R than for ESC) among females
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.95, t-test, 2 sided — This is the test of effect modification by age group; Mean Difference (Final Values) = 1.41, 95% CI 2-sided [-43.38 to 46.20] — A positive value would reflect a larger treatment effect among younger participants compared to older participants
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney) — This is the test of effect modification by viral suppression status; Mean Difference (Final Values) = 5.59, 95% CI 2-sided [-40.47 to 51.65] — A positive value would reflect a greater treatment effect among those with suppressed viral load compared to those without viral suppression
Statistical Analysis 4: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.42, t-test, 2 sided — This is the test of effect modification by QIDS-SR level at entry; Mean Difference (Final Values) = -15.97, 95% CI 2-sided [-58.88 to 26.94] — A negative value would reflect a greater treatment effect among those with moderate depression symptomatology at entry compared to those with severe depression
Statistical Analysis 5: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.68, t-test, 2 sided — This is the test of effect modification by mode of transmission; Mean Difference (Final Values) = 9.99, 95% CI 2-sided [-41.24 to 61.22] — A positive value would reflect a greater treatment effect among those with perinatal transmission compared to behavioral transmission
Statistical Analysis 6: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.57, t-test, 2 sided — This is the test of effect modification by HIV CDC stage; Mean Difference (Final Values) = -14.21, 95% CI 2-sided [-70.62 to 42.20] — A positive value would reflect a greater treatment response among those with HIV CDC Stage 3 classification compared to those with less than Stage 3 classification
Statistical Analysis 7: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.26, t-test, 2 sided — This is the test of effect modification by CD4 Stage; Mean Difference (Final Values) = -44.97, 95% CI 2-sided [-141.12 to 51.17] — A negative value would reflect a greater treatment effect among those with less than Stage 3 CD4 levels compared to those with Stage 3 CD4
Statistical Analysis 8: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.72, t-test, 2 sided — This is the test of effect modification by CD4 nadir stage; Mean Difference (Final Values) = 9.53, 95% CI 2-sided [-52.97 to 72.02] — A positive value would reflect a greater treatment effect by those with Stage 3 CD4 Nadir compared to those with less than Stage 3

21. Secondary Outcome: Behavioral Risk Outcomes: Alcohol Use - Ever Used
Description: The percent of participants who reported ever using alcohol was computed for each site. These site-level percentages were compared across treatment groups.
Time Frame: Weeks 24 and 48
Population: All participants responding to the behavioral risk questionnaire at either week 24 or 48
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 69 | 69
Number analyzed (site) | 6 | 7
percent
  week 24: number analyzed (Participants) | 67 | 69
  week 24 | 75.8 [59.1 to 92.5] | 66.0 [53.0 to 79.0]
  week 48: number analyzed (Participants) | 69 | 60
  week 48 | 70.4 [38.9 to 100.00] | 76.6 [57.8 to 95.5]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The percent of participants with alcohol use ever at week 24 were computed for each site. These site-level percentages were compared across treatment groups; Test type: Superiority; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = 9.9, 95% CI 2-sided [-8.4 to 28.1] — A positive value would indicate site-level percentages were higher in the COMB-R group and vice versa
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; The percent of participants with alcohol use ever at week 48 were computed for each site. These site-level percentages were compared across treatment groups; Test type: Superiority; p = 0.66, t-test, 2 sided; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-37.1 to 24.6] — A positive value would indicate site-level percentages were higher in the COMB-R group and vice versa

22. Secondary Outcome: Behavioral Risk- Alcohol Use - Past 3 Months Regular Use Frequency
Description: Frequency of alcohol use during the past three months was reported for those participants reporting at least some use ever; frequency was measured on a 5-point Likert scale from 1 to 5 (1=Never, 2=Once or twice, 3 = monthly, 4=weekly, 5 = daily or almost daily). A lower score indicates less alcohol use. The percentage of participants at each site with regular use (3=monthly, 4=weekly, 5=daily) was computed. The site-level percentages were compared across treatments.
Time Frame: weeks 24 and 48
Population: All participants with behavior risk responses at week 24 or 48 who also responded that they had used alcohol.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 50 | 46
Number analyzed (site) | 6 | 7
percent
  week 24 | 37.0 [16.5 to 57.6] | 32.3 [10.3 to 54.4]
  week 48: number analyzed (Participants) | 49 | 42
  week 48 | 56.9 [39.0 to 74.7] | 30.2 [0.0 to 60.6]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The percent of participants with regular frequency alcohol use at week 24 were computed for each site. These site-level percentages were compared across treatment groups; Test type: Superiority; p = 0.71, t-test, 2 sided; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-22.3 to 31.7] — A positive value indicates higher site-level percentages in the COMB-R group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; The percent of participants at each site with regular alcohol use at week 48 was computed. These site-level percents were compared across treatments; Test type: Superiority; p = 0.10, t-test, 2 sided; Mean Difference (Final Values) = 26.7, 95% CI 2-sided [-6.3 to 59.6] — A positive value would indicate higher site-level percentages in the COMB-R group

23. Secondary Outcome: Behavioral Risk - Alcohol Use - Number of Drinks Per Day
Description: The number of alcoholic drinks per day on a typical day was reported. The average of the number of drinks for all participants at each site was computed and these site-level averages were compared across treatments. Analysis was limited to those participants reporting at least some use ever.
Time Frame: weeks 24 and 48
Population: All participants with behavior risk data at week 24 or 48 who said they had used alcohol
Measure: Mean (95% Confidence Interval); unit: drinks
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 51 | 47
Number analyzed (site) | 6 | 7
drinks
  week 24 | 1.7 [1.2 to 2.1] | 2.8 [1.4 to 4.2]
  week 48: number analyzed (Participants) | 49 | 42
  week 48 | 2.1 [1.7 to 2.4] | 1.9 [1.1 to 2.8]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The average number of drinks per day reported at week 24 was computed for each site and these site-level averages were compared across treatments; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.6 to 0.2] — A positive value would indicate site level averages were higher in the COMB-R group and vice versa
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; The site-level average numbers of drinks per day reported at week 48 were computed and these site-level averages were compared across treatment groups; Test type: Superiority; p = 0.79, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.8 to 1.0] — A positive value would indicate site level averages were higher in the COMB-R group and vice versa

24. Secondary Outcome: Behavioral Risk - Alcohol Use - Binge Drinking
Description: Binge drinking is defined by the number of days with 5 or more drinks in a row (within a couple of hours) during the past 3 months. These numbers were averaged for all participants at each site and the site-level averages were compared across treatments.Analysis was limited to those participants reporting at least some use ever.
Time Frame: Weeks 24 and 48
Population: All participants with behavior risk responses at week 24 or 48 who also said that they had used alcohol.
Measure: Mean (95% Confidence Interval); unit: days
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 51 | 46
Number analyzed (site) | 6 | 7
days
  week 24 | 1.0 [0.7 to 1.3] | 1.1 [0.2 to 1.9]
  week 48: number analyzed (Participants) | 49 | 42
  week 48 | 0.8 [0.2 to 1.4] | 0.8 [0.2 to 1.4]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The site-level average number of days with binge drinking at week 24 were computed and these site-level averages were compared across treatments; Test type: Superiority; p = 0.87, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.9 to 0.8] — A positive value would indicate site level averages were higher in the COMB-R group anc vice versa
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; The site-level average number of days with binge drinking reported at week 48 were computed and the site-level averages were compared across treatment groups; Test type: Superiority; p = 0.99, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.8 to 0.8] — A positive difference would indicate site level averages were higher in the COMB-R group and vice versa

25. Secondary Outcome: Behavioral Risk Outcomes: Tobacco Use- Ever Used
Description: The percent of participants reporting tobacco use (ever) was computed for each site and these site-level averages were compared across treatments.
Time Frame: Weeks 24 and 48
Population: All participants with behavior risk data at either week 24 or 48.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 70 | 68
Number analyzed (site) | 6 | 7
percent
  week 24: number analyzed (Participants) | 68 | 68
  week 24 | 42.5 [26.1 to 58.9] | 39.3 [20.0 to 58.6]
  week 48: number analyzed (Participants) | 70 | 63
  week 48 | 48.8 [33.0 to 64.6] | 34.1 [13.5 to 54.7]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The percent of participants with tobacco use ever at week 24 were computed for each site. These site-level percentages were compared across treatment groups; Test type: Superiority; p = 0.77, t-test, 2 sided; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [-19.7 to 26.0] — A positive value would indicate site-level percentages were higher in the COMB-R group and vice versa
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; The percent of participants with tobacco use ever at week 48 were computed for each site. These site-level percentages were compared across treatment groups; Test type: Superiority; p = 0.20, t-test, 2 sided; Mean Difference (Final Values) = 14.7, 95% CI 2-sided [-8.9 to 38.4] — A positive value would indicate site-level percentages were higher in the COMB-R group

26. Secondary Outcome: Behavioral Risk - Tobacco Use - Past 3 Months Regular Use Frequency
Description: Past three months frequency of tobacco use was measured on a 5-point Likert scale (1=never, 2=once or twice, 3=monthly, 4 = weekly, 5=daily/almost daily). The percentage of participants with regular use (monthly, weekly or daily) was computed. Analysis was limited to those participants reporting at least some use ever.
Time Frame: weeks 24 and 48
Population: All participants with behavior risk data at weeks 24 or 48 who said that they had used tobacco.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 35 | 28
Number analyzed (site) | 6 | 7
percent
  week 24: number analyzed (Participants) | 29 | 28
  week 24 | 65.4 [55.3 to 75.5] | 50.2 [32.0 to 68.4]
  week 48: number analyzed (Participants) | 35 | 24
  week 48 | 62.3 [34.5 to 90.1] | 41.7 [12.9 to 70.4]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of regular use of tobacco at week 24. The percent of participants at each site with regular use was computed. These site-level percentages were compared across treatment groups; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = 15.2, 95% CI 2-sided [-2.8 to 33.3] — A positive difference would indicate the site level percentages were higher in the COMB-R group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of regular frequency use of tobacco at week 48. Site level percentages of the numbers of participants with regular tobacco use were computed and compared across treatment groups; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = 20.6, 95% CI 2-sided [-14.0 to 55.3] — A positive difference indicates site-level percentages were higher in the COMB-R group

27. Secondary Outcome: Behavioral Risk Outcomes: Drug Use - Ever Used
Description: For each of the following substances (cannabis, cocaine, amphetamine, inhalants, sedatives, hallucinogens, opioids) we computed the percent of participants at each site who reported ever using the substance. We also computed the site-level percentages of participants ever using any illegal substance excluding cannabis.
Time Frame: Weeks 24 and 48
Population: All participants with behavior risk data at weeks 24 and 48.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 70 | 70
Number analyzed (site) | 6 | 7
percent
  Cannabis, week 24: number analyzed (Participants) | 66 | 68
  Cannabis, week 24 | 70.1 [54.5 to 85.7] | 62.2 [45.6 to 78.8]
  Cannabis, week 48: number analyzed (Participants) | 68 | 64
  Cannabis, week 48 | 69.2 [45.4 to 93.0] | 56.2 [41.1 to 71.3]
  Any illegal substance excluding cannabis, week 24: number analyzed (Participants) | 68 | 70
  Any illegal substance excluding cannabis, week 24 | 19.8 [6.3 to 33.3] | 15.1 [0.0 to 38.1]
  Any illegal substance excluding cannabis, week 48: number analyzed (Participants) | 70 | 65
  Any illegal substance excluding cannabis, week 48 | 18.7 [4.7 to 32.6] | 19.3 [0.0 to 41.3]
  Cocaine, week 24: number analyzed (Participants) | 68 | 69
  Cocaine, week 24 | 9.1 [0.0 to 23.9] | 9.0 [0.0 to 25.2]
  Cocaine, week 48: number analyzed (Participants) | 70 | 64
  Cocaine, week 48 | 7.3 [0.0 to 19.7] | 11.0 [0.0 to 31.8]
  Amphetamines, week 24: number analyzed (Participants) | 68 | 67
  Amphetamines, week 24 | 8.9 [8.1 to 9.7] | 7.0 [0.0 to 18.2]
  Amphetamines, week 48: number analyzed (Participants) | 69 | 65
  Amphetamines, week 48 | 5.7 [0.0 to 13.3] | 7.5 [0.0 to 18.0]
  Inhalant, week 24: number analyzed (Participants) | 68 | 68
  Inhalant, week 24 | 3.0 [0.0 to 8.0] | 1.1 [0.0 to 3.8]
  Inhalant, week 48: number analyzed (Participants) | 70 | 65
  Inhalant, week 48 | 2.9 [0.0 to 7.6] | 3.8 [0.0 to 10.7]
  Sedative, week 24: number analyzed (Participants) | 68 | 69
  Sedative, week 24 | 7.7 [0.5 to 15.0] | 4.2 [0.0 to 9.6]
  Sedative, week 48: number analyzed (Participants) | 70 | 65
  Sedative, week 48 | 3.2 [0.0 to 8.4] | 6.8 [0.0 to 15.9]
  Hallucinogen, week 24: number analyzed (Participants) | 68 | 68
  Hallucinogen, week 24 | 4.7 [0.0 to 12.8] | 5.5 [0.0 to 18.9]
  Hallucinogen, week 48: number analyzed (Participants) | 70 | 65
  Hallucinogen, week 48 | 5.9 [0.0 to 13.7] | 8.2 [0.0 to 25.4]
  Opioid, week 24: number analyzed (Participants) | 68 | 69
  Opioid, week 24 | 5.8 [0.0 to 17.3] | 3.2 [0.0 to 8.6]
  Opioid, week 48: number analyzed (Participants) | 70 | 65
  Opioid, week 48 | 3.0 [0.0 to 8.0] | 6.0 [0.0 to 12.6]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The site-level percentages of participants ever using marijuana (cannabis) reported at week 24 were computed and compared across treatment groups; Test type: Superiority; p = 0.41, t-test, 2 sided; Mean Difference (Final Values) = 7.9, 95% CI 2-sided [-12.4 to 28.3] — A positive value would indicate higher site-level percentages in the COMB-R group and vice versa
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; The site-level percentages of participants ever using marijuana (cannabis) reported at week 48 were computed and compared across treatment groups; Test type: Superiority; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = 13.0, 95% CI 2-sided [-10.9 to 36.8] — A positive value would indicate higher site-level percentages in the COMB-R group and vice versa
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; The site-level percentages of participants ever using any illegal substance excluding marijuana (cannabis) reported at week 24 were computed and compared across treatment groups; Test type: Superiority; p = 0.69, t-test, 2 sided; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-20.2 to 29.5] — A positive difference would indicate higher site-level percentages in the COMB-R group and vice versa
Statistical Analysis 4: Comparison: COMB-R vs Enhanced Standard of Care; The site-level percentages of participants ever using any illegal substance excluding marijuana (cannabis) reported at week 48 were computed and compared across treatment groups; Test type: Superiority; p = 0.96, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-24.8 to 23.5] — A positive difference would indicate higher site-level percentages in the COMB-R group and vice versa

28. Secondary Outcome: Behavioral Risk - Drug Use - Past 3 Months Regular Frequency of Use
Description: Past three months use frequency for cannabis, cocaine, amphetamine, inhalants, sedatives, hallucinogens, opioids was assessed. This was measured on a 5-point Likert scale from 1=Never to 5=almost daily. A lower score indicates less frequent use. Scores were dichotomized as regular use (3=monthly, 4=weekly, 5=daily/almost daily) or low use (1=never, 2=once or twice). The percent of participants who used a substance at regularly, given they ever used it, was computed for each site. We also defined a variable of regular frequency of use for any illegal substance, excluding cannabis.
Time Frame: week 24 and 48
Population: We analyzed data for all participants with substance use data reported at either week 24 or week 48. Note that the overall number of participants analyzed includes cannabis use.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 46 | 45
Number analyzed (site) | 6 | 7
percent
  Cannabis, week 24 | 57.3 [37.0 to 77.6] | 47.2 [16.4 to 77.9]
  Cannabis, week 48: number analyzed (Participants) | 46 | 38
  Cannabis, week 48: number analyzed (site) | 6 | 6
  Cannabis, week 48 | 64.9 [42.8 to 87.0] | 65.0 [31.2 to 98.8]
  any illegal substance, excluding cannabis, week 24: number analyzed (Participants) | 13 | 13
  any illegal substance, excluding cannabis, week 24: number analyzed (site) | 6 | 4
  any illegal substance, excluding cannabis, week 24 | 27.8 [0.0 to 68.7] | 3.1 [0.0 to 13.1]
  any illegal substance, excluding cannabis, week 48: number analyzed (Participants) | 13 | 14
  any illegal substance, excluding cannabis, week 48: number analyzed (site) | 5 | 5
  any illegal substance, excluding cannabis, week 48 | 18.3 [0.0 to 54.5] | 36.7 [2.7 to 70.7]
  cocaine, week 24: number analyzed (Participants) | 6 | 7
  cocaine, week 24: number analyzed (site) | 2 | 2
  cocaine, week 24 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  cocaine, week 48: number analyzed (Participants) | 5 | 7
  cocaine, week 48: number analyzed (site) | 2 | 2
  cocaine, week 48 | 25.0 [0.0 to 100.0] | 0.0 [0.0 to 0.0]
  amphetamine, week 24: number analyzed (Participants) | 6 | 6
  amphetamine, week 24: number analyzed (site) | 6 | 3
  amphetamine, week 24 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  amphetamine, week 48: number analyzed (Participants) | 4 | 5
  amphetamine, week 48: number analyzed (site) | 3 | 3
  amphetamine, week 48 | 0.0 [0.0 to 0.0] | 44.4 [0.0 to 100.0]
  inhalant, week 24: number analyzed (Participants) | 2 | 1
  inhalant, week 24: number analyzed (site) | 2 | 1
  inhalant, week 24 | 50.0 [0.0 to 100.0] | 0.0 [lower limit NA] — There is only one observation in this group
  inhalant, week 48: number analyzed (Participants) | 2 | 3
  inhalant, week 48: number analyzed (site) | 2 | 2
  inhalant, week 48 | 50.0 [0.0 to 100.0] | 0.0 [0.0 to 0.0]
  sedative, week 24: number analyzed (Participants) | 5 | 4
  sedative, week 24: number analyzed (site) | 4 | 3
  sedative, week 24 | 50.0 [0.0 to 100.0] | 16.7 [0.0 to 88.4]
  sedative, week 48: number analyzed (Participants) | 2 | 6
  sedative, week 48: number analyzed (site) | 2 | 3
  sedative, week 48 | 50.0 [0.0 to 100.0] | 55.6 [0.0 to 100.0]
  hallucinogen, week 24: number analyzed (Participants) | 3 | 5
  hallucinogen, week 24: number analyzed (site) | 2 | 1
  hallucinogen, week 24 | 0.0 [0.0 to 0.0] | 0.0 [lower limit NA] — There is only one observation in this group
  hallucinogen, week 48: number analyzed (Participants) | 4 | 6
  hallucinogen, week 48: number analyzed (site) | 3 | 2
  hallucinogen, week 48 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  opioid, week 24: number analyzed (Participants) | 4 | 3
  opioid, week 24: number analyzed (site) | 2 | 2
  opioid, week 24 | 0.0 [0.0 to 0.0] | 25.0 [0.0 to 100.0]
  opioid, week 48: number analyzed (Participants) | 2 | 5
  opioid, week 48: number analyzed (site) | 2 | 4
  opioid, week 48 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for regular use of marijuana (cannabis) at week 24. The percent of participants at each site reporting regular use (of those reporting any use) was computed. These site-level percentages were averaged and compared across treatments; Test type: Superiority; p = 0.53, t-test, 2 sided; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [-23.9 to 44.1] — A positive difference indicates a higher site-level percentage of participants reporting regular use fof marijuana in the COMB-R group compared to the ESC group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of regular use of marijuana (cannabis) at week 48. Of those reporting ever used, the percent at each site reporting regular use was computed. These site-level percentages were averaged and compared across treatment groups; Test type: Superiority; p = 1.0, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-35.1 to 34.9] — A positive difference would indicate higher site-level percentages of regular use of marijuana (cannabis) in the COMB-R group compared to the ESC group
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of regular use of any illegal substance, excluding cannabis, at week 24. Of those reporting ever used, the percent at each site reporting regular use was computed. These site-level percentages were averaged and compared across treatment groups; Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 24.7, 95% CI 2-sided [-16.2 to 65.5] — A positive difference would indicate higher site-level percentages of regular substance use in the COMB-R group compared to the ESC group
Statistical Analysis 4: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of regular use of any illegal substance, excluding cannabis, at week 48. Of those reporting ever used, the percent at each site reporting regular use was computed. These site-level percentages were averaged and compared across treatment groups; Test type: Superiority; p = 0.34, t-test, 2 sided; Mean Difference (Final Values) = -18.3, 95% CI 2-sided [-59.5 to 22.9] — [estimate comment as in outcome 28, analysis 3]

29. Secondary Outcome: Behavioral Risk Outcomes: Sex-Risk Behaviors - Sex as Exchange Commodity
Description: We considered a report of sex as exchange commodity if participant reported either that they gave sex in exchange for money, drugs or shelter or if they bought sex with money, drugs or shelter. This was only reported for participants who said they had had some sex (oral, vaginal or anal) ever. The percent of participants at each site who used sex as an exchange commodity was computed and the site-level percentages were compared across treatments.
Time Frame: Weeks 24 and 48
Population: We analyzed data for all participants who had reported they had ever had sex and with behavioral risk data reported at weeks 24 or 48.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 54 | 55
Number analyzed (site) | 6 | 7
percent
  week 24: number analyzed (Participants) | 53 | 55
  week 24 | 31.6 [2.8 to 60.5] | 18.2 [4.7 to 31.7]
  week 48: number analyzed (Participants) | 54 | 47
  week 48 | 24.2 [2.8 to 45.6] | 20.4 [8.1 to 32.8]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for week 24. The percentage of participants at a site who reported using sex as a commodity was calculated and the site-level percentages were averaged and compared across treatments; Test type: Superiority; p = 0.29, t-test, 2 sided; Mean Difference (Final Values) = 13.4, 95% CI 2-sided [-12.9 to 39.6] — A positive value would indicate higher site-level percents in the COMB-R group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for week 48. The percentage of participants at a site who reported using sex as a commodity was calculated and the site-level percentages were averaged and compared across treatments; Test type: Superiority; p = 0.70, t-test, 2 sided; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-17.0 to 24.5] — A positive difference would indicate site-level percentages were higher in the COMB-R group

30. Secondary Outcome: Behavioral Risk Outcomes: Sex-Risk Behaviors - Importance of Using Condom
Description: Participant reported importance that participant or partner use a condom on a scale from 0 to 100 with 0=not important at all, 50= about as important as the other things in my life and 100=most important thing in my life.This was only reported for participants who said they had had some sex (oral, vaginal or anal) ever. The average scores were computed for all participants at each site and the site-level averages were compared across treatments.
Time Frame: weeks 24 and 48
Population: We analyzed data for all participants reporting ever having had sex and with behavioral risk data at weeks 24 or 48.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 54 | 55
Number analyzed (site) | 6 | 7
units on a scale
  week 24: number analyzed (Participants) | 53 | 55
  week 24 | 83.6 [74.6 to 92.5] | 80.7 [65.4 to 96.0]
  week 48: number analyzed (Participants) | 54 | 47
  week 48 | 80.2 [69.1 to 91.3] | 84.9 [75.3 to 94.5]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for week 24. Scores were averaged by site and the site-level averages were averaged and compared across treatment groups; Test type: Superiority; p = 0.71, t-test, 2 sided; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-13.7 to 19.4] — A positive difference indicates the site-level averages were higher for the COMB-R group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for week 48. Scores were averaged by site and the site-level averages were averaged and compared across treatment groups; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-17.5 to 8.1] — A positive value would indicate site-level averages were higher in the COMB-R group

31. Secondary Outcome: Behavioral Risk- Sex Risk Behaviors - Confidence in Condom Use
Description: Participant reports how confident they are that she/he or partner will use condoms. Reported on a scale from 0-100 with 0=I do not think I will use condoms, 50=I have a 50% chance of using a condom; 100=I think I will definitely use a condom.This was only reported for participants who said they had had some sex (oral, vaginal or anal) ever. The average scores were computed for all participants at each site and the site-level averages were compared across treatments.
Time Frame: Week 24 and 48
Population: We analyzed data for everyone who reported having ever had sex and with behavior risk data at weeks 24 or 48.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 54 | 55
Number analyzed (site) | 6 | 7
units on a scale
  week 24: number analyzed (Participants) | 53 | 55
  week 24 | 78.0 [68.2 to 87.8] | 70.7 [60.6 to 80.8]
  week 48: number analyzed (Participants) | 54 | 46
  week 48 | 78.4 [68.7 to 88.1] | 80.8 [67.5 to 94.1]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 30, analysis 1]; Test type: Superiority; p = 0.23, t-test, 2 sided; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [-5.3 to 19.8] — A positive value would indicate site-level averages were higher in the COMB-R group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; [analysis description as in outcome 30, analysis 2]; Test type: Superiority; p = 0.73, t-test, 2 sided; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-17.5 to 12.7] — A positive difference would indicate site-level averages were higher in the COMB-R group

32. Secondary Outcome: Behavioral Risk - Sex Risk Behaviors - Number of Sexual Partners in Past Three Months
Description: The participant reported the number of sexual partners in the past three months. This was only reported for participants who said they had had some sex (oral, vaginal or anal) ever. The average number of sexual partners was computed for all participants at each site and the site-level summaries were compared across treatment groups.
Time Frame: week 24 and 48
Population: We analyzed data for all participants who reported ever having had sex and who had data at weeks 24 or 48.
Measure: Mean (95% Confidence Interval); unit: partners
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 54 | 55
Number analyzed (site) | 6 | 7
partners
  week 24: number analyzed (Participants) | 53 | 55
  week 24 | 1.9 [0.9 to 2.8] | 1.4 [0.8 to 1.9]
  week 48: number analyzed (Participants) | 54 | 47
  week 48 | 1.6 [1.0 to 2.1] | 1.2 [0.7 to 1.7]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for week 24. Numbers of partners were averaged by site and the site-level averages were averaged and compared across treatment groups; Test type: Superiority; p = 0.24, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.4 to 1.5] — A positive value would indicate site-level averages were higher in COMB-R group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for week 48. Numbers of partners were averaged by site and the site-level averages were averaged and compared across treatment groups; Test type: Superiority; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.3 to 1.0] — A positive difference indicates site-level averages were higher in the COMB-R group

33. Secondary Outcome: Behavioral Risk - Sex Risk Behaviors. Low Use Frequency of Condom Use in Last Three Months - Main Partner
Description: Main partner frequency of condom use was measured on a 5-point Likert scale from 1= always, 2 = more than half the time, 3= about half the time, 4=less than half the time to 5=never. It is only reported if participant reported some anal or vaginal sex in past three months. The worse (higher) score of that reported for vaginal or anal sex is analyzed. For each site we computed the percent of participants reporting low frequency of condom use (score = 3, 4 or 5). The site-level percentages were averaged and the site-level averages were compared across treatments.
Time Frame: week 24 and 48
Population: We analyzed data for all participants reporting one or more sexual partner in past 3 months with data at week 24 or 48 and who reported vaginal or anal sex.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 37 | 35
Number analyzed (site) | 6 | 7
percent
  week 24 | 31.9 [18.9 to 44.8] | 40.1 [8.5 to 71.8]
  week 48: number analyzed (Participants) | 37 | 32
  week 48 | 26.4 [8.8 to 44.1] | 48.2 [19.5 to 76.9]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for week 24 data. We computed the percent of participants reporting low frequency of condom use in past three months by site, averaged the site-level percents and compared these averages across treatment arms; Test type: Superiority; p = 0.57, t-test, 2 sided; Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-40.4 to 23.9] — A positive value would indicate higher site-level percents of low frequency condom use in COMB-R treatment group and vice versa
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for week 48 data. We computed the percent of participants reporting low frequency of condom use in past three months by site, averaged the site-level percents and compared these averages across treatment arms; Test type: Superiority; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = -21.8, 95% CI 2-sided [-53.1 to 9.5] — A positive difference would indicate higher site-level percentages in the COMB-R group and vice versa

34. Secondary Outcome: Behavioral Risk - Sex Risk Behavior - Low Use Frequency of Condom Use in Past 3 Months - Other Partner
Description: Condom use frequency for other than main partners was measured on a 5-point Likert scale from 1= always, 2 = more than half the time, 3= about half the time, 4=less than half the time to 5=never. It is only reported if participant reported some anal or vaginal sex in past three months. The worse (higher) score of that reported for vaginal or anal sex is analyzed. For each site we computed the percent of participants reporting low frequency of condom use (score = 3, 4 or 5). The site-level percentages were averaged and the site-level averages were compared across treatments.
Time Frame: week 24 and 48
Population: We analyzed data for all participants reporting one or more sexual partner in past 3 months and who reported either anal or vaginal sex, with data from weeks 24 or 48.
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 33 | 25
Number analyzed (site) | 6 | 7
percent
  week 24: number analyzed (Participants) | 29 | 25
  week 24 | 28.9 [16.9 to 40.9] | 35.7 [2.0 to 69.4]
  week 48: number analyzed (Participants) | 33 | 23
  week 48 | 14.4 [0.0 to 30.9] | 52.1 [22.3 to 82.0]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; We computed the site-level percentages of participants reporting low frequency condom use at week 24, then averaged the site-level percentages by treatment group and compared these group average percents; Test type: Superiority; p = 0.65, t-test, 2 sided; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-40.9 to 27.2] — A positive difference would indicate site level percents were higher in the COMB-R group and vice versa
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; We computed the site-level percentages of participants reporting low frequency condom use at week 48, then averaged the site-level percentages by treatment group and compared these group average percents; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = -37.8, 95% CI 2-sided [-69.7 to -5.8] — A positive difference would indicate site-level percentages were higher in the COMB-R group and vice versa

35. Secondary Outcome: To Describe the Implementation Fidelity at COMB-R Sites and the Counseling Strategies and Medication Patterns at ESC Sites: The Total Numbers of Counseling Sessions
Description: We counted the total numbers of COMB-R and ESC counseling sessions administered over the intervention period (through week 24), including both interim and scheduled visits. The average number of sessions was computed for all participants at each site and those averages were compared across treatments.
Time Frame: over 24 weeks
Population: We analyzed data for all study participants
Measure: Mean (95% Confidence Interval); unit: sessions
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 81 | 75
Number analyzed (site) | 6 | 7
sessions | 11.5 [9.3 to 13.7] | 9.0 [3.5 to 14.4]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; We averaged the number of counseling sessions for each site and compared these site-level averages; Test type: Superiority; p = 0.33, t-test, 2 sided; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-3.0 to 8.1] — A positive difference indicates COMB-R participants attended more sessions than ESC

36. Secondary Outcome: Implementation Fidelity (COMB-R Sites) - Count of Participants Having Been Administered Various COMB-R Counseling Approaches
Description: For COMB-R; we assessed numbers of participants for whom counselors reported using each type of cognitive behavioral therapy (CBT) approaches over the intervention period. A participant was counted in a specific category if the approach was ever used during the 24 week intervention period.
Time Frame: over 24 Weeks
Population: We analyzed data for all COMB-R participants with at least one counseling session over the 24 week treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | COMB-R
Number analyzed (Participants) | 80
Participants
  Psychoeducation | 80
  Motivational interviewing | 77
  Adherence training | 63
  Behavioral coping | 79
  Cognitive restructuring | 70
  Problem solving | 68
  Wellness | 74
  Practice and application | 75
  Homework assignment | 76
  Relapse and wellness plan | 59
  Safety plan | 38
  Booster sessions | 26
  Family communication | 40
  Contingency management | 19
  Emotional regulation | 53

37. Secondary Outcome: Counseling Strategies (ESC Sites) - Count of Participants Having Been Administered Various ESC Counseling Approaches
Description: We summarized the types of counseling approaches used by the ESC clinicians over the intervention period. A participant was counted in a specific category if the approach was ever used during the 24 week intervention period.
Time Frame: Over 24 weeks
Population: We analyzed all participants in the ESC group with at least one counseling session.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Standard of Care
Number analyzed (Participants) | 75
Participants
  Supportive/coping with stress | 47
  Cognitive behavioral | 35
  Focused problem solving | 24
  Interpersonal | 15
  Expressive or emotion focused | 12
  Motivational interviewing or enhancement | 12
  Eclectic or personalized treatment | 7
  Other | 5
  Acceptance and commitment | 2
  Dialectical behavioral | 2
  Relaxation and/or mindfulness | 2
  Substance use focused treatment | 1

38. Secondary Outcome: Implementation Fidelity (COMB-R Sites); Medication Management - Number of Sessions
Description: We computed the number of Medication Management (MM) sessions attended by participants in the COMB-R group over 24 weeks including both interim and scheduled visits .We averaged the number of sessions for all participants at each site and then took the mean of the site-level averages.
Time Frame: Over 24 Weeks
Population: We analyzed data for all COMB-R study participants
Measure: Mean (Standard Deviation); unit: sessions
Units Other Than Participants: site
Arm/Group | COMB-R
Number analyzed (Participants) | 81
Number analyzed (site) | 6
sessions | 5.3 (2.2)

39. Secondary Outcome: Implemental Fidelity (COMB-R) - Medication Management - Stages
Description: We summarized the stages of the MM algorithm reported for participants by prescribing clinicians in the COMB-R group. Stage 0 is no medication. Stage 1 is monotherapy with a selective serotonin re-uptake inhibitor (SSRI). Stage 2 is monotherapy with a second SSRI. Stage 3 is monotherapy with a non-SSRI. Stage 4 is combination treatment with two antidepressants or an antidepressant plus lithium. Stages 1 through 3 also allow for partial responders to receive augmentation with selected other psychiatric medications.
Time Frame: week 1, 6, 12, 24
Population: We analyzed data for all COMB-R participants with a medication management session administered.
Measure: Count of Participants; unit: Participants
Arm/Group | COMB-R
Number analyzed (Participants) | 78
Participants
  week 1: Stage 0 | 54
  week 1: Stage 1 | 19
  week 1: Stage 2 | 1
  week 1: Stage 3 | 4
  week 6: number analyzed (Participants) | 73
  week 6: Stage 0 | 46
  week 6: Stage 1 | 22
  week 6: Stage 2 | 1
  week 6: Stage 3 | 4
  week 12: number analyzed (Participants) | 71
  week 12: Stage 0 | 45
  week 12: Stage 1 | 20
  week 12: Stage 2 | 3
  week 12: Stage 3 | 3
  week 24: number analyzed (Participants) | 69
  week 24: Stage 0 | 38
  week 24: Stage 1 | 25
  week 24: Stage 2 | 3
  week 24: Stage 3 | 3

40. Secondary Outcome: Acceptability: Frequency of Psychiatric Medication Use - Percent of Participants on Psychiatric Medications
Description: We assessed whether or not participants were taking psychiatric medications at week 24 and we computed the percent of participants at each site taking psychiatric medications overall and by classes of psychiatric medications. We compared the site-level percentages across treatment groups. Classes of medications included: any psychiatric medication, any antidepressant medication, any regimen with a selective serotonin re uptake inhibitor (SSRI), any regimen with a non-SSRI antidepressant medication, any other non-antidepressant psychiatric medication.
Time Frame: week 24
Population: We analyzed all participants on study at week 24
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 74 | 72
Number analyzed (site) | 6 | 7
percent
  Any psychiatric medications | 49.1 [40.1 to 58.0] | 30.4 [11.7 to 49.1]
  Any antidepressant medication | 44.9 [34.7 to 55.1] | 27.5 [10.9 to 44.2]
  SSRI | 40.7 [26.9 to 54.6] | 18.4 [3.5 to 33.2]
  non-SSRI | 6.4 [0.0 to 14.2] | 10.3 [0.0 to 22.5]
  Other non-antidepressant psychiatric medication | 10.1 [0.0 to 21.4] | 15.1 [0.0 to 33.9]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis for the percent of participants on any psychiatric medication at week 24. Site-level percentages were compared across treatments; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = 18.7, 95% CI 2-sided [-0.9 to 38.2] — A positive difference indicates more participants in the COMB-R group were taking medications, based on site-level percentages
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of the percent of participants on antidepressant medications. Site-level percentages were compared across treatments; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [-0.7 to 35.5] — A positive difference means the site-level percentages of those taking medications were higher in the COMB-R group
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of the percent of participants on SSRI antidepressant medications. Site-level percentages were compared across treatments; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = 22.4, 95% CI 2-sided [4.2 to 40.6] — A positive difference indicates the site-level percentages of those taking medications were higher in the COMB-R group
Statistical Analysis 4: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of the percent of participants on non-SSRI antidepressant medications. Site-level percentages were compared across treatments; Test type: Superiority; p = 0.54, t-test, 2 sided; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-17.3 to 9.6] — A positive difference would indicate site-level percentages of those on medication were higher in the COMB-R group
Statistical Analysis 5: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of the percent of participants on non-antidepressant psychiatric medications. Site-level percentages were compared across treatments; Test type: Superiority; p = 0.60, t-test, 2 sided; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-25.4 to 15.4] — A positive value would indicate the site-level percentages of those on medications were higher in the COMB-R group

41. Secondary Outcome: Acceptability - Frequency of Psychiatric Medication Use - Percent of Study Time on Psychiatric Medications Through Week 24
Description: For those participants taking each of several classes of psychiatric medications during the first 24 study weeks, we computed the percent of study time during which each participant was taking psychiatric medications of that category. Regimen classes were: any psychiatric medication, any antidepressant medication, single selective serotonin re-uptake inhibitor (SSRI), single non-SSRI, SSRI+other medication, non-SSRI+other medication. Then the average percent of time on each category of medication was computed for all participants at each site. The site-level means were compared across treatments.
Time Frame: over 24 weeks
Population: For each class of psychiatric medication, participants who had received it at some time during the first 24 weeks of the study.
Measure: Mean (95% Confidence Interval); unit: percentage of time on medication
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 44 | 27
Number analyzed (site) | 6 | 7
percentage of time on medication
  any psychiatric medication | 69.3 [50.0 to 88.5] | 73.1 [48.3 to 97.9]
  Single SSRI: number analyzed (Participants) | 33 | 7
  Single SSRI: number analyzed (site) | 6 | 5
  Single SSRI | 60.9 [46.3 to 75.5] | 62.8 [18.6 to 106.9]
  SSRI+other: number analyzed (Participants) | 11 | 8
  SSRI+other: number analyzed (site) | 5 | 5
  SSRI+other | 39.2 [7.5 to 70.8] | 55.8 [14.0 to 97.7]
  single non-SSRI: number analyzed (Participants) | 3 | 7
  single non-SSRI: number analyzed (site) | 2 | 5
  single non-SSRI | 59.1 [58.2 to 59.9] | 72.5 [19.0 to 126.1]
  non-SSRI plus other: number analyzed (Participants) | 2 | 5
  non-SSRI plus other: number analyzed (site) | 2 | 1
  non-SSRI plus other | 64.5 [-386.9 to 515.9] | 60.6 [lower limit NA] — Only one site had data
  Any antidepressant: number analyzed (Participants) | 40 | 24
  Any antidepressant | 69.8 [53.6 to 85.9] | 74.0 [49.3 to 98.6]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis comparing site-level mean percents of study time on any psychiatric medication across treatment groups; Test type: Superiority; p = 0.77, t-test, 2 sided; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-32.5 to 24.8] — A positive difference would indicate more time on medication in the COMB-R group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis comparing site-level mean percents of study time on single SSRI psychiatric medication across treatment groups; Test type: Superiority; p = 0.91, t-test, 2 sided; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-37.3 to 33.5] — A positive difference would indicate more study time on medication in the COMB-R group
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis comparing site-level mean percents of study time on SSRI+other psychiatric medication across treatment groups; Test type: Superiority; p = 0.40, t-test, 2 sided; Mean Difference (Final Values) = -16.7, 95% CI 2-sided [-60.2 to 26.9] — A positive value would indicate more time on medication in the COMB-R group
Statistical Analysis 4: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis comparing site-level mean percents of study time on a single non-SSRI psychiatric medication across treatment groups; Test type: Superiority; p = 0.52, t-test, 2 sided; Mean Difference (Final Values) = -13.5, 95% CI 2-sided [-67.0 to 40.1] — A positive difference would indicate more time on medication in COMB-R group
Statistical Analysis 5: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis comparing site-level mean percents of study time on non-SSRI+other psychiatric medication across treatment groups. This analysis is unstable because of sparseness; Test type: Superiority; p = 0.96, t-test, 2 sided; Because of sparseness, the confidence intervals for this site-level analysis are very large; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-778.0 to 785.7] — A positive difference indicates more time on medication in the COMB-R group. There was data from only one site in the ESC group and 2 sites in the COMB-R group. The confidence interval for the difference is quite large and the test is unreliable
Statistical Analysis 6: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis comparing site-level mean percents of study time on antidepressant medication across treatment groups; Test type: Superiority; p = 0.74, t-test, 2 sided; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-31.4 to 23.0] — A positive difference would reflect more time on medications in the COMB-R group

42. Secondary Outcome: Acceptability: Number of Interim Visits - Counseling Sessions
Description: We counted the number of interim visits with the counseling clinician, defined as those outside of the scheduled study visits. The average number for all participants at each site were computed. Site mean numbers were compared across treatments.
Time Frame: Over 24 Weeks
Population: We analyzed data for all study participants
Measure: Mean (95% Confidence Interval); unit: sessions
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 81 | 75
Number analyzed (site) | 6 | 7
sessions | 7.9 [5.7 to 10.2] | 5.3 [-0.1 to 10.7]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; We compared the site-level average number of interim counseling sessions between treatment groups; Test type: Superiority; p = 0.29, t-test, 2 sided; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-2.8 to 8.2] — A positive difference would indicate the site level average interim counseling sessions was higher in the COMB-R group

43. Secondary Outcome: Acceptability - Number of Interim Medication Management Visits (COMB-R)
Description: We counted the number of interim visits with the prescribing clinician, defined as those outside of the scheduled study visits. We computed the average number of sessions for all participants at each site. We took the mean of those averages.
Time Frame: Over 24 weeks
Population: We analyzed data for all COMB-R participants
Measure: Mean (Standard Deviation); unit: sessions
Units Other Than Participants: site
Arm/Group | COMB-R
Number analyzed (Participants) | 81
Number analyzed (site) | 6
sessions | 1.7 (2.1)

44. Secondary Outcome: COMB-R and ESC Acceptability Among Participants
Description: Client satisfaction was computed as the mean of the 8 questionnaire items. Each is rated on a 4-point Likert scale from 1-4, with 4 being the best acceptability. Items reflected quality of service, degree to which program met participant needs, and satisfaction with and efficacy of the help given. The average score for all participants at each site was computed. Site mean scores were compared across treatments.
Time Frame: Week 24
Population: All participants with at least one counseling clinician, prescribing clinician or participant acceptability questionnaire completed
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 68 | 70
Number analyzed (site) | 6 | 7
units on a scale | 3.67 [3.52 to 3.81] | 3.47 [3.32 to 3.61]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The average score for all participants at each site was computed. These site-level averages were compared across treatment groups; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [0.02 to 0.38] — A positive difference indicates higher site-level averages in the COMB-R group

45. Secondary Outcome: COMB-R and ESC Acceptability Among Counseling Clinicians
Description: Six items were rated on a 4-point Likert scale from 0-3 (0=poor, 1=fair, 2=good, 3=excellent). A higher score indicates better clinician satisfaction with administering the intervention. These questions rated appropriateness, effectiveness, flexibility, ease of use, fit and overall quality of the treatment approach. For each participant's clinician, a mean score of the six items was computed. The average score was computed for the clinicians of all participants at each site. These site-level means were compared between groups.
Time Frame: Week 24
Population: as for outcome 44
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 68 | 71
Number analyzed (site) | 6 | 7
units on a scale | 2.26 [1.90 to 2.62] | 2.33 [2.10 to 2.56]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The average of scores for all participants' clinicians at each site was computed and these site-level averages were compared across treatments; Test type: Superiority; p = 0.69, t-test, 2 sided; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.43 to 0.29] — A positive difference would indicate the site-level averages were higher in the COMB-R group compared to the ESC group and vice versa

46. Secondary Outcome: COMB-R MM and ESC Acceptability Among Prescribing Clinicians
Description: For each participant's prescribing clinician, we assessed two domains: How easy or difficult it was to follow the treatment plan (ESC) or medication management algorithm (COMB-R) and whether or not participants symptoms improved over the intervention period. These items were assessed on a 5-point Likert scale (0, 1, 2, 3, 4) and reverse scored if necessary so that a higher score reflected that it was easier to follow the algorithm and that the patients' symptoms improved. Average scores at each site were computed and the site-level summaries were compared across treatments.
Time Frame: Week 24
Population: Prescribing clinician responses for all participants with at least one counseling clinician, prescribing clinician or participant acceptability questionnaire completed. For the ESC group, prescribing clinicians sometimes did not complete the questions if participant was not on medication for depression.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 69 | 40
Number analyzed (site) | 6 | 7
units on a scale | 3.05 [2.73 to 3.37] | 2.40 [2.10 to 2.70]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; The average scores for all participants' prescribing clinicians at each site were computed and these site-level averages were compared across treatment groups; Test type: Superiority; p = 0.004, t-test, 2 sided; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [0.26 to 1.03] — A positive difference would indicate site-level averages were higher for the COMB-R group than the ESC group and vice versa

47. Secondary Outcome: Grade 3 or Higher Adverse Events (AE), Psychological Hospitalizations, and Suicide Attempts
Description: In this analysis only "new" events were counted; as identified by MedDRA Preferred Term; that is, those which were first reported after study entry. Two types of adverse events were reported: 1) grade 3 or higher signs/symptoms, and 2) grade 3 or higher diagnoses. "Trigger" events (psychiatric hospitalization or suicide attempts) were also reported. For each of these three types of events, the percent of participants at each site with at least one such event was computed. The average of these site-level percentages within each treatment arm were compared. Note, in some cases due to sparseness (few events reported at sites within a treatment group), the lower bound of the 95% confidence interval was less than zero . In those cases, the bounds were truncated to zero.
Time Frame: Over 24 Weeks
Population: This is the analysis for the Week 24 data. We count a participant if any new qualifying event was reported prior to the week 24 upper window (+30 days).
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 81 | 75
Number analyzed (site) | 6 | 7
percent
  Week 24, Mean % with Grade 3+ signs/symptoms | 9.27 [2.40 to 16.14] | 9.11 [0.0 to 22.53]
  Week 24, Mean % with Grade 3+ diagnoses | 10.48 [1.56 to 19.40] | 7.92 [0.05 to 15.79]
  Week 24, Mean % with AE trigger event | 5.59 [0.0 to 13.18] | 1.19 [0.0 to 4.10]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of new Grade 3+ signs/symptoms through week 24. The percent of participants at each site with at least one such event was computed. The average of these site-level percents was calculated for each treatment arm. These averages were compared; Test type: Superiority — We tested the null hypothesis that the treatment group means were equal vs. not; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-14.04 to 14.36] — We subtract group mean for ESC from group mean for COMB-R. The group means are the means of the site-level percentages of participants with events
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of new Grade 3+ diagnoses through week 24.The percent of participants at each site with at least one such event was computed. The average of these site-level percents was calculated for each treatment arm. These averages were compared; Test type: Superiority — We tested the null hypothesis that the treatment group means were equal vs. not; p = 0.60, t-test, 2 sided; Mean Difference (Final Values) = 2.57, 95% CI 2-sided [-7.85 to 12.98] — We subtracted the group mean for the ESC group from that of the COMB-R group. The group mean is the mean of the site-specific percentages of participants with events
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of the triggering events (psychiatric hospitalizations or suicide attempts) through week 24. A participant is counted once if they had reported any such event prior to the upper bound of the week 24 window. The percent of participants at each site with at least one such event were computed.The average of these site-level percents was calculated for each treatment arm. These averages were compared; Test type: Superiority — We tested the null hypothesis that the treatment group means were equal vs. not.The group mean is the mean of the site-specific percentages of participants with events as defined above; p = 0.17, t-test, 2 sided; Mean Difference (Final Values) = 4.40, 95% CI 2-sided [-2.21 to 11.02] — The ESC group mean percent of participants reporting a trigger event was subtracted from the COMB-R group mean

48. Secondary Outcome: Grade 3 or Higher Adverse Events (AE), Psychological Hospitalizations, and Suicide Attempts
Description: n this analysis only "new" events were counted; as identified by MedDRA Preferred Term; that is, those which were first reported after study entry. Two types of adverse events were reported: 1) grade 3 or higher signs/symptoms, and 2) grade 3 or higher diagnoses. "Trigger" events (psychiatric hospitalization or suicide attempts) were also reported. For each of these three types of events, the percent of participants at each site with at least one such event was computed. The average of these site-level percentages within each treatment arm were compared. Note, in some cases due to sparseness (few events reported at sites within a treatment group), the lower bound of the 95% confidence interval was less than zero . In those cases, the bounds were truncated to zero.
Time Frame: Over 48 weeks
Population: This is the analysis for the Week 48 data. We count a participant if any new qualifying event was reported prior to the week 48 upper window (+30 days).
Measure: Mean (95% Confidence Interval); unit: percent
Units Other Than Participants: site
Arm/Group | COMB-R | Enhanced Standard of Care
Number analyzed (Participants) | 81 | 75
Number analyzed (site) | 6 | 7
percent
  Week 48, Mean % with Grade 3+ sign/symptoms | 13.12 [4.35 to 21.88] | 12.98 [0.52 to 25.43]
  Week 48, Mean % with Grade 3+ diagnoses | 19.22 [5.81 to 32.62] | 13.57 [3.77 to 23.37]
  Week 48, Mean % with AE trigger event | 6.88 [0.00 to 15.56] | 3.87 [0.00 to 8.64]
Statistical Analysis 1: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of new Grade 3+ signs/symptoms through week 48. The percent of participants at each site with at least one such event was computed. The average of these site-level percents was calculated for each treatment arm. These averages were compared; Test type: Superiority; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-13.85 to 14.13] — A positive difference indicates more participants with events in the COMB-R group
Statistical Analysis 2: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of new Grade 3+ diagnoses through week 48. The percent of participants at each site with at least one such event was computed. The average of these site-level percents was calculated for each treatment arm. These averages were compared; Test type: Superiority; p = 0.40, t-test, 2 sided; Mean Difference (Final Values) = 5.64, 95% CI 2-sided [-8.60 to 19.89] — A positive difference indicates more participants with events in the COMB-R group
Statistical Analysis 3: Comparison: COMB-R vs Enhanced Standard of Care; This is the analysis of new trigger events through week 48. The percent of participants at each site with at least one such event was computed. The average of these site-level percents was calculated for each treatment arm. These averages were compared; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = 3.01, 95% CI 2-sided [-5.27 to 11.29] — A positive difference indicates more participants with events in the COMB-R group

ADVERSE EVENTS:
Time Frame: The adverse event data were collected over the 48 weeks of the study duration.
Description: At entry, all diagnoses and signs/symptoms occurring within 30 days of entry were collected. Post-entry, all new diagnoses and signs/symptoms of ≥Grade 3 were collected. Laboratory events related to an adverse event or hospitalization were collected. Suicide attempts and psychological hospitalizations were also collected. The Division of AIDS (DAIDS) AE Grading Table (Corrected version 2.1) and EAE Manual (V2.0) were used. All eligible participants who initiated study treatment are included.
Groups:
- Enhanced Standard of Care (ESC): Ongoing psychopharmacological and psychosocial counseling and treatment for depression at HIV clinical treatment centers enhanced by providing clinicians with up-to-date information and didactic training.
Arm/Group | COMB-R | Enhanced Standard of Care (ESC)
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/75
Serious Adverse Events (participants affected / at risk) | 6/81 | 6/75
Other Adverse Events (participants affected / at risk) | 50/81 | 49/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COMB-R (N=81) | Enhanced Standard of Care (ESC) (N=75)
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 3 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | COMB-R (N=81) | Enhanced Standard of Care (ESC) (N=75)
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Fatigue (General disorders) | 1 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4
Disturbance in attention (Nervous system disorders) | 0 | 10
Lethargy (Nervous system disorders) | 0 | 8
Anxiety (Psychiatric disorders) | 5 | 2
Depressed mood (Psychiatric disorders) | 3 | 11
Depression (Psychiatric disorders) | 25 | 12
Insomnia (Psychiatric disorders) | 1 | 10
Irritability (Psychiatric disorders) | 0 | 11
Major depression (Psychiatric disorders) | 22 | 25
Persistent depressive disorder (Psychiatric disorders) | 7 | 10
Suicidal ideation (Psychiatric disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02939131/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT02939131/Prot_ICF_001.pdf